CLINICAL TRIAL: NCT03814590
Title: Phase I/II, Observer-blind, Safety, Reactogenicity and Immunogenicity Study of GSK Biologicals' Respiratory Syncytial Virus (RSV) Vaccine GSK3844766A in Subjects Aged 18-40 or 60-80 Years
Brief Title: A Study to Assess the Safety, Reactogenicity and Immune Response of GlaxoSmithKline (GSK) Biologicals' Investigational Respiratory Syncytial Virus (RSV) Vaccine (GSK3844766A) in Older Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 208851; 2018-000849-38 (EudraCT Number)
Record Dates: First submitted 2019-01-11; First posted 2019-01-24 (Actual); Results first posted 2022-03-23 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-07

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus (RSV); Vaccine; Safety; Reactogenicity; Immunogenicity
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Respiratory Syncytial Virus Vaccines; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Group Low Dose_PLAIN_A (Experimental): Subjects in Part A, aged 18-40 years, receiving 2 doses of RSV Vaccine (GSK3844766A) unadjuvanted low dose on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Biological: RSV Vaccine (GSK3844766A) unadjuvanted low dose
- Group Medium Dose_PLAIN_A (Experimental): Subjects in Part A aged 18-40 years, receiving 2 doses of RSV Vaccine (GSK3844766A) unadjuvanted medium dose, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Biological: RSV Vaccine (GSK3844766A) unadjuvanted medium dose
- Group High Dose_PLAIN_A (Experimental): Subjects in Part A aged 18-40 years, receiving 2 doses of RSV Vaccine (GSK3844766A) unadjuvanted high dose, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Biological: RSV Vaccine (GSK3844766A) unadjuvanted high dose
- Group Placebo_A (Placebo Comparator): Subjects in Part A aged 18-40 years, receiving 2 doses of placebo (saline solution) control, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Drug: Placebo (Saline solution)
- Group Low Dose_PLAIN_B (Experimental): Subjects in Part B aged 60-80 years, receiving 2 doses of RSV Vaccine (GSK3844766A) unadjuvanted low dose, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Biological: RSV Vaccine (GSK3844766A) unadjuvanted low dose
- Group Low Dose_AS01E_B (Experimental): Subjects in Part B aged 60-80 years, receiving 2 doses of the RSV Vaccine (GSK3844766A) low dose adjuvanted with AS01E, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Biological: RSV Vaccine (GSK3844766A) low dose adjuvanted with AS01E
- Group Low Dose_AS01B_B (Experimental): Subjects in Part B aged 60-80 years, receiving 2 doses of the RSV Vaccine (GSK3844766A) low dose adjuvanted with AS01B, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Biological: RSV Vaccine (GSK3844766A) low dose adjuvanted with AS01B
- Group Medium Dose_PLAIN_B (Experimental): Subjects in Part B aged 60-80 years, receiving 2 doses of RSV Vaccine (GSK3844766A) unadjuvanted medium dose, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Biological: RSV Vaccine (GSK3844766A) unadjuvanted medium dose
- Group Medium Dose_AS01E_B (Experimental): Subjects in Part B aged 60-80 years, receiving 2 doses of the RSV Vaccine (GSK3844766A) medium dose adjuvanted with AS01E, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Biological: RSV Vaccine (GSK3844766A) medium dose adjuvanted with AS01E
- Group Medium Dose_AS01B_B (Experimental): Subjects in Part B aged 60-80 years, receiving 2 doses of the RSV Vaccine (GSK3844766A) medium dose adjuvanted with AS01B, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Biological: RSV Vaccine (GSK3844766A) medium dose adjuvanted with AS01B
- Group High Dose_PLAIN_B (Experimental): Subjects in Part B aged 60-80 years, receiving 2 doses of RSV Vaccine (GSK3844766A) unadjuvanted high dose, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Biological: RSV Vaccine (GSK3844766A) unadjuvanted high dose
- Group High Dose_AS01E_B (Experimental): Subjects in Part B aged 60-80 years, receiving 2 doses of the RSV Vaccine (GSK3844766A) high dose adjuvanted with AS01E, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Biological: RSV Vaccine (GSK3844766A) high dose adjuvanted with AS01E
- Group High Dose_AS01B_B (Experimental): Subjects in Part B aged 60-80 years, receiving 2 doses of the RSV Vaccine (GSK3844766A) high dose adjuvanted with AS01B, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Biological: RSV Vaccine (GSK3844766A) high dose adjuvanted with AS01B
- Group Placebo_B (Placebo Comparator): Subjects in Part B aged 60-80 years, receiving 2 doses of placebo (saline solution) control, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
  Interventions: Drug: Placebo (Saline solution)

INTERVENTIONS:
Biological: RSV Vaccine (GSK3844766A) unadjuvanted low dose — Two doses administered intramuscularly at Days 1 and 61 in the deltoid region of the arm
  Arms: Group Low Dose_PLAIN_A; Group Low Dose_PLAIN_B
Biological: RSV Vaccine (GSK3844766A) low dose adjuvanted with AS01E — Two doses administered intramuscularly at Days 1 and 61 in the deltoid region of the arm.
  Arms: Group Low Dose_AS01E_B
Biological: RSV Vaccine (GSK3844766A) low dose adjuvanted with AS01B — Two doses administered intramuscularly at Days 1 and 61 in the deltoid region of the arm
  Arms: Group Low Dose_AS01B_B
Biological: RSV Vaccine (GSK3844766A) unadjuvanted medium dose — Two doses administered intramuscularly at Days 1 and 61 in the deltoid region of the arm.
  Arms: Group Medium Dose_PLAIN_A; Group Medium Dose_PLAIN_B
Biological: RSV Vaccine (GSK3844766A) medium dose adjuvanted with AS01E — Two doses administered intramuscularly at Days 1 and 61 in the deltoid region of the arm.
  Arms: Group Medium Dose_AS01E_B
Biological: RSV Vaccine (GSK3844766A) medium dose adjuvanted with AS01B — Two doses administered intramuscularly at Days 1 and 61 in the deltoid region of the arm.
  Arms: Group Medium Dose_AS01B_B
Biological: RSV Vaccine (GSK3844766A) unadjuvanted high dose — Two doses administered intramuscularly at Days 1 and 61 in the deltoid region of the arm.
  Arms: Group High Dose_PLAIN_A; Group High Dose_PLAIN_B
Biological: RSV Vaccine (GSK3844766A) high dose adjuvanted with AS01E — Two doses administered intramuscularly at Days 1 and 61 in the deltoid region of the arm
  Arms: Group High Dose_AS01E_B
Biological: RSV Vaccine (GSK3844766A) high dose adjuvanted with AS01B — Two doses administered intramuscularly at Days 1 and 61 in the deltoid region of the arm.
  Arms: Group High Dose_AS01B_B
Drug: Placebo (Saline solution) — Two doses administered intramuscularly at Days 1 and 61 in the deltoid region of the arm.
  Arms: Group Placebo_A; Group Placebo_B

SUMMARY:
The purpose of this study is to assess the safety, reactogenicity and immune responses of two doses of the investigational RSV vaccines (with different formulations), when administered intramuscularly (IM) according to a 0, 2 month schedule, in older adults aged 60 to 80 years.

As the investigational vaccines have not yet been tested in humans before, the study will first assess the safety, reactogenicity and immune responses in young adults aged 18 to 40 years. The study will thus be conducted in 2 parts (Part A and Part B).

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performing any study specific procedure.

For Part A:

• A male or female between, and including, 18 and 40 years of age at the time of the first vaccination.

For Part B:

* A male or female between, and including, 60 and 80 years of age at the time of the first vaccination.
* Subjects with residence status allowing free mixing with general community or in an assisted-living facility that provides minimal assistance, such that the subject is primarily responsible for self-care and activities of daily living.

Exclusion Criteria:

For all subjects:

* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before the first dose of study vaccine, or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make IM injection unsafe.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting 6 months prior to the first vaccine dose. For corticosteroids, this will mean prednisone (≥ 20 mg/day, or equivalent). Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs or planned administration at any time during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of study vaccine administration, with the exception of inactivated and subunit influenza vaccines which can be administered up to 14 days before or from 30 days after each study vaccination.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to latex.
* Serious or unstable chronic illness. Patients with chronic stable conditions with or without specific treatment, such as diabetes, hypertension or cardiac disease, are allowed to participate in this study.
* Any other condition (e.g. chronic obstructive pulmonary disease or severe respiratory condition) that, in the opinion of the investigator, might interfere with the evaluations required by the study.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by the investigator based on medical history, physical examination or laboratory screening tests.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the first dose of study vaccine or planned administration during the study period.
* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.
* Previous vaccination with an RSV vaccine.
* Lymphoproliferative disorder and malignancy within 5 years.
* Body mass index > 40 kg/m².
* Planned move to a location that will prohibit participating in the trial until study end.
* At screening: Hematology parameters (complete blood cell count [red blood cells, white blood cells], white blood cells differential count [lymphocytes, neutrophils and eosinophils], platelets count or hemoglobin level) and/or biochemistry parameters (creatinine, blood urea nitrogen or liver enzymes [alanine aminotransferase or aspartate aminotransferase]) outside the normal laboratory ranges, unless the laboratory abnormalities are considered not clinically significant by the investigator.

For Part A:

* Pregnant or lactating female.
* Female subjects of childbearing potential, except if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

For Part B:

* Known previous administration of a vaccine containing MPL, QS-21 and/or MF59 (e.g. GSK Biologicals' vaccine against human papillomavirus infection marketed as Cervarix, GSK Biologicals' Herpes Zoster vaccine marketed as Shingrix, an adjuvanted recombinant varicella zoster virus envelope gE subunit vaccine [HZ/su], or MF59 adjuvanted influenza vaccines [e.g. Fluad]).
* Planned administration of GSK Biologicals' Herpes Zoster vaccine marketed as Shingrix or an adjuvanted recombinant varicella zoster virus envelope gE subunit vaccine [HZ/su] within 180 days after the second dose of the study vaccine.
* Bedridden subjects.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (21):
- United States (18):
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Lenexa, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Elkridge, Maryland
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Hickory, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
- Belgium (3):
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Wilrijk

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Leroux-Roels I, Davis MG, Steenackers K, Essink B, Vandermeulen C, Fogarty C, Andrews CP, Kerwin E, David MP, Fissette L, Vanden Abeele C, Collete D, de Heusch M, Salaun B, De Schrevel N, Koch J, Verheust C, Dezutter N, Struyf F, Mesaros N, Tica J, Hulstrom V. Safety and Immunogenicity of a Respiratory Syncytial Virus Prefusion F (RSVPreF3) Candidate Vaccine in Older Adults: Phase 1/2 Randomized Clinical Trial. J Infect Dis. 2023 Mar 28;227(6):761-772. doi: 10.1093/infdis/jiac327. PMID 35904987

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1053 participants received the study vaccine or placebo and were included in the Exposed Set.
Groups:
- Low Dose_PLAIN_A Group: Subjects in Part A, aged 18-40 years, receiving 2 doses of RSV Vaccine (GSK3844766A) unadjuvanted low dose, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
- Medium Dose_PLAIN_A Group: Subjects in Part A aged 18-40 years, receiving 2 doses of RSV Vaccine (GSK3844766A) unadjuvanted medium dose, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
- High Dose_PLAIN_A Group: Subjects in Part A aged 18-40 years, receiving 2 doses of RSV Vaccine (GSK3844766A) unadjuvanted high dose, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
- Placebo_A Group: Subjects in Part A aged 18-40 years, receiving 2 doses of placebo (Saline solution) control, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
- Low Dose_PLAIN_B Group: Subjects in Part B aged 60-80 years, receiving 2 doses of RSV Vaccine (GSK3844766A) unadjuvanted low dose, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
- Medium Dose_PLAIN_B Group: Subjects in Part B aged 60-80 years, receiving 2 doses of RSV Vaccine (GSK3844766A) unadjuvanted medium dose, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
- High Dose_PLAIN_B Group: Subjects in Part B aged 60-80 years, receiving 2 doses of RSV Vaccine (GSK3844766A) unadjuvanted high dose, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
- Low Dose_AS01E_B Group: Subjects in Part B aged 60-80 years, receiving 2 doses of the RSV Vaccine (GSK3844766A) low dose adjuvanted with AS01E, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
- Medium Dose_AS01E_B Group: Subjects in Part B aged 60-80 years, receiving 2 doses of the RSV Vaccine (GSK3844766A) medium dose adjuvanted with AS01E, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
- High Dose_AS01E_B Group: Subjects in Part B aged 60-80 years, receiving 2 doses of the RSV Vaccine (GSK3844766A) high dose adjuvanted with AS01E, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
- Low Dose_AS01B_B Group: Subjects in Part B aged 60-80 years, receiving 2 doses of the RSV Vaccine (GSK3844766A) low dose adjuvanted with AS01B, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
- Medium Dose_AS01B_B Group: Subjects in Part B aged 60-80 years, receiving 2 doses of the RSV Vaccine (GSK3844766A) medium dose adjuvanted with AS01B, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
- High Dose_AS01B_B Group: Subjects in Part B aged 60-80 years, receiving 2 doses of the RSV Vaccine (GSK3844766A) high dose adjuvanted with AS01B, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
- Placebo_B Group: Subjects in Part B aged 60-80 years, receiving 2 doses of placebo (Saline solution) control, on a 0, 2 Months schedule, by IM injection into the deltoid region of the arm.
Period: Overall Study
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Started | 12 | 12 | 12 | 12 | 101 | 97 | 100 | 101 | 101 | 100 | 103 | 100 | 101 | 101
Completed | 12 | 10 | 11 | 12 | 100 | 92 | 97 | 95 | 101 | 95 | 100 | 100 | 97 | 98
Not Completed | 0 | 2 | 1 | 0 | 1 | 5 | 3 | 6 | 0 | 5 | 3 | 0 | 4 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 3 | 0
Not completed — Lost to Follow-up | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — CONSENT WITHDRAWAL, DUE TO COVID-19 BUT NOT DUE TO AN ADVERSE EVENT | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — CONSENT WITHDRAWAL, NOT DUE TO COVID-19 AND NOT DUE TO AN ADVERSE EVENT | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 3 | 1 | 0 | 1 | 2
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — UNKNOWN REASON | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 101 | 97 | 100 | 101 | 101 | 100 | 103 | 100 | 101 | 101 | 1053
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.2 (7.0) | 26.5 (4.0) | 29.9 (6.1) | 31.6 (5.6) | 67.3 (5.6) | 67.8 (5.6) | 67.9 (4.9) | 67.8 (5.1) | 67.1 (5.6) | 67.6 (5.2) | 67.6 (4.9) | 67.5 (4.9) | 67.5 (4.9) | 68.1 (5.7) | 65.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 7 | 9 | 58 | 54 | 57 | 58 | 57 | 57 | 59 | 58 | 57 | 58 | 604
  Male | 4 | 5 | 5 | 3 | 43 | 43 | 43 | 43 | 44 | 43 | 44 | 42 | 44 | 43 | 449
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  ASIAN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  BLACK OR AFRICAN AMERICAN | 2 | 1 | 2 | 1 | 5 | 7 | 4 | 12 | 7 | 5 | 11 | 7 | 7 | 4 | 75
  OTHER | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 5
  WHITE | 10 | 10 | 10 | 11 | 95 | 90 | 93 | 88 | 94 | 93 | 92 | 93 | 92 | 97 | 968

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Solicited Local Symptoms After First Vaccination Dose
Description: Assessed solicited local AEs at injection site are pain, erythema and swelling. Any erythema/swelling was scored as injection site erythema/swelling with a diameter larger than (>) 20 millimeters (mm)
Time Frame: During a 7-day follow-up period after first vaccination dose (i.e., on the day of vaccination [at Day 1] and 6 subsequent days)
Population: The analysis was performed on the Exposed Set that includes all subjects with at least one study vaccine administration documented and with the subject diary completed after the first vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 12 | 12 | 11 | 12 | 100 | 96 | 99 | 101 | 100 | 100 | 103 | 99 | 101 | 98
Participants
  Erythema | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 5 | 6 | 9 | 16 | 15 | 18 | 1
  Pain | 1 | 7 | 6 | 0 | 9 | 5 | 14 | 54 | 57 | 56 | 78 | 63 | 76 | 4
  Swelling | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 7 | 7 | 6 | 10 | 7 | 9 | 0

2. Primary Outcome: Number of Subjects With Any Solicited Local Symptoms After Second Vaccination Dose
Description: as for outcome 1
Time Frame: During a 7-day follow-up period after second vaccination dose (i.e., on the day of vaccination [at Day 61] and 6 subsequent days)
Population: The analysis was performed on the Exposed Set that includes all subjects with at least one study vaccine administration documented and with the subject diary completed after the second vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 12 | 10 | 11 | 12 | 95 | 91 | 90 | 94 | 94 | 95 | 96 | 93 | 93 | 97
Participants
  Erythema | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 3 | 3 | 7 | 16 | 14 | 12 | 0
  Pain | 5 | 7 | 8 | 1 | 18 | 18 | 23 | 34 | 48 | 47 | 58 | 56 | 59 | 4
  Swelling | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3 | 3 | 6 | 10 | 7 | 10 | 0

3. Primary Outcome: Number of Subjects With Any Solicited General Symptom After First Vaccination Dose
Description: Assessed solicited general symptoms include arthralgia, fatigue, fever [defined as temperature equal to or above 38.0 degrees Celsius (°C)], gastrointestinal symptoms [nausea, vomiting, diarrhea and/or abdominal pain], headache, myalgia and shivering.
Time Frame: During a 7-day follow-up period after the first vaccination dose (i.e., on the day of vaccination [at Day 1] and 6 subsequent days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 12 | 12 | 11 | 12 | 100 | 96 | 99 | 101 | 100 | 100 | 103 | 99 | 101 | 98
Participants
  Arthralgia | 0 | 0 | 0 | 0 | 7 | 4 | 0 | 7 | 12 | 6 | 15 | 9 | 17 | 7
  Fatigue | 4 | 5 | 1 | 6 | 22 | 11 | 24 | 26 | 28 | 21 | 30 | 29 | 49 | 16
  Fever | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 1 | 3 | 3 | 1 | 0
  Gastrointestinal symptoms | 1 | 2 | 1 | 1 | 8 | 8 | 10 | 8 | 8 | 9 | 13 | 7 | 13 | 10
  Headache | 2 | 4 | 3 | 2 | 8 | 7 | 13 | 20 | 12 | 17 | 28 | 27 | 28 | 8
  Myalgia | 0 | 1 | 1 | 0 | 4 | 3 | 1 | 9 | 8 | 6 | 19 | 12 | 18 | 5
  Shivering | 0 | 2 | 0 | 1 | 1 | 1 | 2 | 6 | 5 | 3 | 12 | 8 | 16 | 1

4. Primary Outcome: Number of Subjects With Any Solicited General Symptom After Second Vaccination Dose
Description: as for outcome 3
Time Frame: During a 7-day follow-up period after the second vaccination dose (i.e., on the day of vaccination [at Day 61] and 6 subsequent days)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 12 | 10 | 11 | 12 | 95 | 91 | 90 | 94 | 94 | 95 | 96 | 93 | 93 | 97
Participants
  Arthralgia | 0 | 0 | 0 | 0 | 1 | 4 | 2 | 8 | 8 | 10 | 21 | 11 | 13 | 4
  Fatigue | 3 | 2 | 4 | 5 | 16 | 11 | 13 | 24 | 22 | 24 | 35 | 35 | 34 | 16
  Fever | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 4 | 6 | 3 | 0
  Gastrointestinal symptoms | 1 | 1 | 2 | 2 | 4 | 2 | 7 | 7 | 5 | 7 | 11 | 7 | 9 | 6
  Headache | 2 | 2 | 3 | 3 | 11 | 9 | 8 | 15 | 18 | 10 | 33 | 26 | 18 | 9
  Myalgia | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 6 | 9 | 11 | 19 | 12 | 18 | 2
  Shivering | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 3 | 4 | 14 | 12 | 9 | 2

5. Primary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) After Any Vaccination Dose
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and/or any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any is defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During a 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) after any vaccination dose (across doses)
Population: The analysis was performed on the Exposed Set that includes all subjects with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 101 | 97 | 100 | 101 | 101 | 100 | 103 | 100 | 101 | 101
Participants | 2 | 4 | 4 | 6 | 34 | 28 | 30 | 40 | 29 | 36 | 39 | 34 | 43 | 33

6. Primary Outcome: Number of Subjects Presenting Change From Baseline in Hematology and Biochemistry With Respect of Normal Laboratory Ranges, After First Vaccine Dose (Part A Groups)
Description: Assessed hematological laboratory parameters include basophils, eosinophils, erythrocytes, hemoglobin, lymphocytes, monocytes, neutrophils, platelets, white blood cells. Biochemical laboratory parameters include alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine, urea nitrogen and uric acid. Categories reported when comparing Day 1 (pre-vaccination dose 1=baseline) and Day 8 hematological and biochemical laboratory results are defined as follows: <parameter>-<range at baseline>-<range at timing> (e.g. ALT-Within-Within). Ranges level being classified as unknown, below, within or above the normal ranges.
Time Frame: At baseline and at 7 days after the first vaccine dose (Day 8)
Population: The analysis was performed on the Exposed Set that includes all subjects from Part A groups, with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group
Number analyzed (Participants) | 12 | 12 | 11 | 12
Participants
  ALT-WITHIN-WITHIN | 12 | 12 | 11 | 12
  AST-WITHIN-WITHIN: number analyzed (Participants) | 11 | 12 | 11 | 11
  AST-WITHIN-WITHIN | 11 | 12 | 11 | 11
  AST-ABOVE-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 1
  AST-ABOVE-WITHIN | 1 | 0 | 0 | 1
  Basophils-WITHIN-WITHIN | 12 | 12 | 11 | 12
  Creatinine-BELOW-BELOW: number analyzed (Participants) | 1 | 2 | 0 | 1
  Creatinine-BELOW-BELOW | 0 | 0 | 0 | 1
  Creatinine-BELOW-WITHIN: number analyzed (Participants) | 1 | 2 | 0 | 1
  Creatinine-BELOW-WITHIN | 1 | 2 | 0 | 0
  Creatinine-WITHIN-WITHIN: number analyzed (Participants) | 11 | 9 | 11 | 11
  Creatinine-WITHIN-WITHIN | 11 | 9 | 11 | 11
  Creatinine-ABOVE-ABOVE: number analyzed (Participants) | 0 | 1 | 0 | 0
  Creatinine-ABOVE-ABOVE | 0 | 1 | 0 | 0
  Eosinophils-BELOW-BELOW: number analyzed (Participants) | 0 | 1 | 1 | 0
  Eosinophils-BELOW-BELOW | 0 | 1 | 0 | 0
  Eosinophils-BELOW-WITHIN: number analyzed (Participants) | 0 | 1 | 1 | 0
  Eosinophils-BELOW-WITHIN | 0 | 0 | 1 | 0
  Eosinophils-WITHIN-WITHIN: number analyzed (Participants) | 11 | 10 | 10 | 12
  Eosinophils-WITHIN-WITHIN | 11 | 10 | 10 | 12
  Eosinophils-ABOVE-WITHIN: number analyzed (Participants) | 1 | 1 | 0 | 0
  Eosinophils-ABOVE-WITHIN | 1 | 1 | 0 | 0
  Erythrocytes-BELOW-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 1
  Erythrocytes-BELOW-WITHIN | 1 | 0 | 0 | 1
  Erythrocytes-WITHIN-WITHIN: number analyzed (Participants) | 11 | 11 | 11 | 11
  Erythrocytes-WITHIN-WITHIN | 11 | 11 | 11 | 11
  Erythrocytes-ABOVE-WITHIN: number analyzed (Participants) | 0 | 1 | 0 | 0
  Erythrocytes-ABOVE-WITHIN | 0 | 1 | 0 | 0
  Hemoglobin-BELOW-BELOW: number analyzed (Participants) | 1 | 0 | 0 | 1
  Hemoglobin-BELOW-BELOW | 0 | 0 | 0 | 1
  Hemoglobin-BELOW-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 1
  Hemoglobin-BELOW-WITHIN | 1 | 0 | 0 | 0
  Hemoglobin-WITHIN-WITHIN: number analyzed (Participants) | 11 | 12 | 11 | 11
  Hemoglobin-WITHIN-WITHIN | 11 | 12 | 11 | 11
  Lymphocytes-BELOW-WITHIN: number analyzed (Participants) | 0 | 1 | 0 | 1
  Lymphocytes-BELOW-WITHIN | 0 | 1 | 0 | 1
  Lymphocytes-WITHIN-WITHIN: number analyzed (Participants) | 12 | 11 | 11 | 11
  Lymphocytes-WITHIN-WITHIN | 12 | 11 | 11 | 11
  Monocytes-BELOW-WITHIN: number analyzed (Participants) | 0 | 1 | 0 | 0
  Monocytes-BELOW-WITHIN | 0 | 1 | 0 | 0
  Monocytes-WITHIN-WITHIN: number analyzed (Participants) | 12 | 11 | 11 | 12
  Monocytes-WITHIN-WITHIN | 12 | 11 | 11 | 12
  Neutrophis-BELOW-BELOW: number analyzed (Participants) | 2 | 1 | 1 | 0
  Neutrophis-BELOW-BELOW | 0 | 0 | 1 | 0
  Neutrophils-BELOW-WITHIN: number analyzed (Participants) | 2 | 1 | 1 | 0
  Neutrophils-BELOW-WITHIN | 2 | 1 | 0 | 0
  Neutrophils-WITHIN-WITHIN: number analyzed (Participants) | 8 | 11 | 10 | 12
  Neutrophils-WITHIN-WITHIN | 8 | 11 | 10 | 12
  Neutrophils-ABOVE-WITHIN: number analyzed (Participants) | 2 | 0 | 0 | 0
  Neutrophils-ABOVE-WITHIN | 1 | 0 | 0 | 0
  Neutrophils-ABOVE-ABOVE: number analyzed (Participants) | 2 | 0 | 0 | 0
  Neutrophils-ABOVE-ABOVE | 1 | 0 | 0 | 0
  Platelets-WITHIN-WITHIN | 12 | 12 | 11 | 12
  Urea Nitrogen-WITHIN-BELOW | 0 | 0 | 0 | 1
  Urea Nitrogen-WITHIN-WITHIN | 12 | 12 | 11 | 11
  Uric Acid-BELOW-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 0
  Uric Acid-BELOW-WITHIN | 1 | 0 | 0 | 0
  Uric Acid-WITHIN-WITHIN: number analyzed (Participants) | 11 | 12 | 11 | 12
  Uric Acid-WITHIN-WITHIN | 11 | 12 | 11 | 12
  White Blood Cells-BELOW-BELOW: number analyzed (Participants) | 2 | 1 | 1 | 1
  White Blood Cells-BELOW-BELOW | 0 | 1 | 0 | 0
  White Blood Cells-BELOW-WITHIN: number analyzed (Participants) | 2 | 1 | 1 | 1
  White Blood Cells-BELOW-WITHIN | 2 | 0 | 1 | 1
  White Blood Cells-WITHIN-WITHIN: number analyzed (Participants) | 8 | 11 | 10 | 11
  White Blood Cells-WITHIN-WITHIN | 8 | 11 | 10 | 11
  White Blood Cells-ABOVE-WITHIN: number analyzed (Participants) | 2 | 0 | 0 | 0
  White Blood Cells-ABOVE-WITHIN | 1 | 0 | 0 | 0
  White Blood Cells-ABOVE-ABOVE: number analyzed (Participants) | 2 | 0 | 0 | 0
  White Blood Cells-ABOVE-ABOVE | 1 | 0 | 0 | 0

7. Primary Outcome: Number of Subjects Presenting Change From Baseline in Hematology and Biochemistry With Respect of Normal Laboratory Ranges, After First Vaccine Dose (Part B Groups)
Description: as for outcome 6
Time Frame: At baseline and at 7 days after the first vaccine dose (Day 8)
Population: The analysis was performed on the Exposed Set that includes all subjects from Part B groups, with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 101 | 97 | 99 | 100 | 100 | 100 | 103 | 100 | 101 | 101
Participants
  ALT-WITHIN-UNKNOWN: number analyzed (Participants) | 100 | 97 | 99 | 98 | 98 | 100 | 100 | 95 | 99 | 100
  ALT-WITHIN-UNKNOWN | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  ALT-WITHIN-WITHIN: number analyzed (Participants) | 100 | 97 | 99 | 98 | 98 | 100 | 100 | 95 | 99 | 100
  ALT-WITHIN-WITHIN | 99 | 97 | 98 | 97 | 98 | 100 | 100 | 94 | 98 | 98
  ALT-WITHIN-ABOVE: number analyzed (Participants) | 100 | 97 | 99 | 98 | 98 | 100 | 100 | 95 | 99 | 100
  ALT-WITHIN-ABOVE | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  ALT-ABOVE-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 2 | 2 | 0 | 3 | 5 | 2 | 1
  ALT-ABOVE-WITHIN | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0 | 0
  ALT-ABOVE-ABOVE: number analyzed (Participants) | 1 | 0 | 0 | 2 | 2 | 0 | 3 | 5 | 2 | 1
  ALT-ABOVE-ABOVE | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 3 | 2 | 1
  AST-WITHIN-UNKNOWN: number analyzed (Participants) | 101 | 97 | 99 | 100 | 99 | 99 | 99 | 98 | 100 | 101
  AST-WITHIN-UNKNOWN | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 1
  AST-WITHIN-WITHIN: number analyzed (Participants) | 101 | 97 | 99 | 100 | 99 | 99 | 99 | 98 | 100 | 101
  AST-WITHIN-WITHIN | 100 | 97 | 98 | 98 | 99 | 98 | 97 | 97 | 98 | 99
  AST-WITHIN-ABOVE: number analyzed (Participants) | 101 | 97 | 99 | 100 | 99 | 99 | 99 | 98 | 100 | 101
  AST-WITHIN-ABOVE | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  AST-ABOVE-WITHIN: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 2 | 1 | 0
  AST-ABOVE-WITHIN | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0
  AST-ABOVE-ABOVE: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 2 | 1 | 0
  AST-ABOVE-ABOVE | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1 | 0
  Basophils-WITHIN-UNKNOWN | 0 | 1 | 0 | 1 | 4 | 2 | 0 | 0 | 0 | 0
  Basophils-WITHIN-WITHIN | 100 | 96 | 99 | 99 | 96 | 98 | 103 | 100 | 101 | 100
  Basophils-WITHIN-ABOVE | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine-BELOW-BELOW: number analyzed (Participants) | 1 | 8 | 6 | 3 | 5 | 2 | 4 | 5 | 5 | 1
  Creatinine-BELOW-BELOW | 0 | 5 | 4 | 3 | 4 | 0 | 1 | 3 | 2 | 0
  Creatinine-BELOW-WITHIN: number analyzed (Participants) | 1 | 8 | 6 | 3 | 5 | 2 | 4 | 5 | 5 | 1
  Creatinine-BELOW-WITHIN | 1 | 3 | 2 | 0 | 1 | 2 | 3 | 2 | 3 | 1
  Creatinine-WITHIN-UNKNOWN: number analyzed (Participants) | 94 | 85 | 92 | 94 | 95 | 95 | 97 | 92 | 94 | 99
  Creatinine-WITHIN-UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Creatinine-WITHIN-BELOW: number analyzed (Participants) | 94 | 85 | 92 | 94 | 95 | 95 | 97 | 92 | 94 | 99
  Creatinine-WITHIN-BELOW | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 5 | 3
  Creatinine-WITHIN-WITHIN: number analyzed (Participants) | 94 | 85 | 92 | 94 | 95 | 95 | 97 | 92 | 94 | 99
  Creatinine-WITHIN-WITHIN | 92 | 83 | 89 | 92 | 92 | 93 | 93 | 90 | 88 | 95
  Creatinine-WITHIN-ABOVE: number analyzed (Participants) | 94 | 85 | 92 | 94 | 95 | 95 | 97 | 92 | 94 | 99
  Creatinine-WITHIN-ABOVE | 1 | 1 | 2 | 1 | 2 | 1 | 3 | 1 | 0 | 0
  Creatinine-ABOVE-UNKNOWN: number analyzed (Participants) | 6 | 4 | 1 | 3 | 0 | 3 | 2 | 3 | 2 | 1
  Creatinine-ABOVE-UNKNOWN | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine-ABOVE-WITHIN: number analyzed (Participants) | 6 | 4 | 1 | 3 | 0 | 3 | 2 | 3 | 2 | 1
  Creatinine-ABOVE-WITHIN | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Creatinine-ABOVE-ABOVE: number analyzed (Participants) | 6 | 4 | 1 | 3 | 0 | 3 | 2 | 3 | 2 | 1
  Creatinine-ABOVE-ABOVE | 4 | 4 | 1 | 1 | 0 | 2 | 2 | 2 | 2 | 1
  Eosinophils-BELOW-BELOW: number analyzed (Participants) | 7 | 6 | 5 | 4 | 4 | 7 | 9 | 6 | 5 | 3
  Eosinophils-BELOW-BELOW | 2 | 3 | 4 | 0 | 3 | 5 | 3 | 4 | 2 | 2
  Eosinophils-BELOW-WITHIN: number analyzed (Participants) | 7 | 6 | 5 | 4 | 4 | 7 | 9 | 6 | 5 | 3
  Eosinophils-BELOW-WITHIN | 5 | 3 | 1 | 3 | 1 | 2 | 5 | 2 | 3 | 1
  Eosinophils-BELOW-ABOVE: number analyzed (Participants) | 7 | 6 | 5 | 4 | 4 | 7 | 9 | 6 | 5 | 3
  Eosinophils-BELOW-ABOVE | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Eosinophils-WITHIN-UNKNOWN: number analyzed (Participants) | 90 | 89 | 90 | 94 | 95 | 92 | 91 | 92 | 94 | 96
  Eosinophils-WITHIN-UNKNOWN | 0 | 1 | 0 | 1 | 4 | 2 | 0 | 0 | 0 | 0
  Eosinophils-WITHIN-BELOW: number analyzed (Participants) | 90 | 89 | 90 | 94 | 95 | 92 | 91 | 92 | 94 | 96
  Eosinophils-WITHIN-BELOW | 3 | 1 | 2 | 2 | 1 | 1 | 3 | 5 | 3 | 5
  Eosinophils-WITHIN-WITHIN: number analyzed (Participants) | 90 | 89 | 90 | 94 | 95 | 92 | 91 | 92 | 94 | 96
  Eosinophils-WITHIN-WITHIN | 85 | 86 | 88 | 91 | 89 | 88 | 88 | 86 | 90 | 90
  Eosinophils-WITHIN-ABOVE: number analyzed (Participants) | 90 | 89 | 90 | 94 | 95 | 92 | 91 | 92 | 94 | 96
  Eosinophils-WITHIN-ABOVE | 2 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1
  Eosinophils-ABOVE-WITHIN: number analyzed (Participants) | 4 | 2 | 4 | 2 | 1 | 1 | 3 | 2 | 2 | 2
  Eosinophils-ABOVE-WITHIN | 2 | 1 | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Eosinophils-ABOVE-ABOVE: number analyzed (Participants) | 4 | 2 | 4 | 2 | 1 | 1 | 3 | 2 | 2 | 2
  Eosinophils-ABOVE-ABOVE | 2 | 1 | 0 | 1 | 1 | 1 | 3 | 2 | 2 | 0
  Erythrocytes-BELOW-BELOW: number analyzed (Participants) | 5 | 4 | 1 | 1 | 4 | 4 | 2 | 1 | 3 | 3
  Erythrocytes-BELOW-BELOW | 4 | 3 | 0 | 1 | 4 | 3 | 2 | 1 | 1 | 2
  Erythrocytes-BELOW-WITHIN: number analyzed (Participants) | 5 | 4 | 1 | 1 | 4 | 4 | 2 | 1 | 3 | 3
  Erythrocytes-BELOW-WITHIN | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 1
  Erythrocytes-WITHIN-UNKNOWN: number analyzed (Participants) | 95 | 91 | 96 | 99 | 95 | 94 | 97 | 98 | 97 | 95
  Erythrocytes-WITHIN-UNKNOWN | 0 | 1 | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 0
  Erythrocytes-WITHIN-BELOW: number analyzed (Participants) | 95 | 91 | 96 | 99 | 95 | 94 | 97 | 98 | 97 | 95
  Erythrocytes-WITHIN-BELOW | 5 | 1 | 0 | 0 | 3 | 3 | 2 | 1 | 4 | 1
  Erythrocytes-WITHIN-WITHIN: number analyzed (Participants) | 95 | 91 | 96 | 99 | 95 | 94 | 97 | 98 | 97 | 95
  Erythrocytes-WITHIN-WITHIN | 89 | 89 | 95 | 98 | 88 | 89 | 95 | 96 | 93 | 94
  Erythrocytes-WITHIN-ABOVE: number analyzed (Participants) | 95 | 91 | 96 | 99 | 95 | 94 | 97 | 98 | 97 | 95
  Erythrocytes-WITHIN-ABOVE | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
  Erythrocytes-ABOVE-WITHIN: number analyzed (Participants) | 1 | 2 | 2 | 0 | 1 | 2 | 4 | 1 | 1 | 3
  Erythrocytes-ABOVE-WITHIN | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 1 | 0
  Erythrocytes-ABOVE-ABOVE: number analyzed (Participants) | 1 | 2 | 2 | 0 | 1 | 2 | 4 | 1 | 1 | 3
  Erythrocytes-ABOVE-ABOVE | 1 | 1 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 3
  Hemoglobin-BELOW-UNKNOWN: number analyzed (Participants) | 10 | 8 | 1 | 5 | 7 | 6 | 4 | 4 | 9 | 2
  Hemoglobin-BELOW-UNKNOWN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin-BELOW-BELOW: number analyzed (Participants) | 10 | 8 | 1 | 5 | 7 | 6 | 4 | 4 | 9 | 2
  Hemoglobin-BELOW-BELOW | 9 | 5 | 1 | 4 | 7 | 4 | 4 | 3 | 5 | 1
  Hemoglobin-BELOW-WITHIN: number analyzed (Participants) | 10 | 8 | 1 | 5 | 7 | 6 | 4 | 4 | 9 | 2
  Hemoglobin-BELOW-WITHIN | 1 | 2 | 0 | 1 | 0 | 2 | 0 | 1 | 4 | 1
  Hemoglobin-WITHIN-UNKNOWN: number analyzed (Participants) | 91 | 86 | 97 | 93 | 92 | 94 | 98 | 95 | 91 | 98
  Hemoglobin-WITHIN-UNKNOWN | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 0
  Hemoglobin-WITHIN-BELOW: number analyzed (Participants) | 91 | 86 | 97 | 93 | 92 | 94 | 98 | 95 | 91 | 98
  Hemoglobin-WITHIN-BELOW | 4 | 3 | 1 | 1 | 1 | 2 | 2 | 3 | 5 | 2
  Hemoglobin-WITHIN-WITHIN: number analyzed (Participants) | 91 | 86 | 97 | 93 | 92 | 94 | 98 | 95 | 91 | 98
  Hemoglobin-WITHIN-WITHIN | 87 | 83 | 96 | 91 | 88 | 90 | 96 | 90 | 86 | 95
  Hemoglobin-WITHIN-ABOVE: number analyzed (Participants) | 91 | 86 | 97 | 93 | 92 | 94 | 98 | 95 | 91 | 98
  Hemoglobin-WITHIN-ABOVE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
  Hemoglobin-ABOVE-WITHIN: number analyzed (Participants) | 0 | 3 | 1 | 2 | 1 | 0 | 1 | 1 | 1 | 1
  Hemoglobin-ABOVE-WITHIN | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1
  Hemoglobin-ABOVE-ABOVE: number analyzed (Participants) | 0 | 3 | 1 | 2 | 1 | 0 | 1 | 1 | 1 | 1
  Hemoglobin-ABOVE-ABOVE | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
  Lymphocytes-BELOW-BELOW: number analyzed (Participants) | 2 | 2 | 0 | 3 | 3 | 3 | 4 | 2 | 1 | 1
  Lymphocytes-BELOW-BELOW | 1 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 1
  Lymphocytes-BELOW-WITHIN: number analyzed (Participants) | 2 | 2 | 0 | 3 | 3 | 3 | 4 | 2 | 1 | 1
  Lymphocytes-BELOW-WITHIN | 1 | 2 | 0 | 2 | 3 | 2 | 2 | 1 | 1 | 0
  Lymphocytes-WITHIN-UNKNOWN: number analyzed (Participants) | 99 | 94 | 99 | 97 | 96 | 97 | 99 | 98 | 100 | 100
  Lymphocytes-WITHIN-UNKNOWN | 0 | 1 | 0 | 1 | 4 | 2 | 0 | 0 | 0 | 0
  Lymphocytes-WITHIN-BELOW: number analyzed (Participants) | 99 | 94 | 99 | 97 | 96 | 97 | 99 | 98 | 100 | 100
  Lymphocytes-WITHIN-BELOW | 0 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 2
  Lymphocytes-WITHIN-WITHIN: number analyzed (Participants) | 99 | 94 | 99 | 97 | 96 | 97 | 99 | 98 | 100 | 100
  Lymphocytes-WITHIN-WITHIN | 99 | 92 | 99 | 94 | 90 | 94 | 96 | 98 | 100 | 98
  Lymphocytes-WITHIN-ABOVE: number analyzed (Participants) | 99 | 94 | 99 | 97 | 96 | 97 | 99 | 98 | 100 | 100
  Lymphocytes-WITHIN-ABOVE | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Lymphocytes-ABOVE-WITHIN: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocytes-ABOVE-WITHIN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes-ABOVE-ABOVE: number analyzed (Participants) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocytes-ABOVE-ABOVE | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Monocytes-BELOW-UNKNOWN: number analyzed (Participants) | 4 | 2 | 3 | 2 | 1 | 4 | 5 | 6 | 4 | 3
  Monocytes-BELOW-UNKNOWN | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Monocytes-BELOW-BELOW: number analyzed (Participants) | 4 | 2 | 3 | 2 | 1 | 4 | 5 | 6 | 4 | 3
  Monocytes-BELOW-BELOW | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 5 | 2 | 0
  Monocytes-BELOW-WITHIN: number analyzed (Participants) | 4 | 2 | 3 | 2 | 1 | 4 | 5 | 6 | 4 | 3
  Monocytes-BELOW-WITHIN | 3 | 1 | 3 | 2 | 0 | 1 | 5 | 1 | 2 | 3
  Monocytes-WITHIN-UNKNOWN: number analyzed (Participants) | 97 | 95 | 96 | 98 | 99 | 96 | 98 | 94 | 97 | 98
  Monocytes-WITHIN-UNKNOWN | 0 | 1 | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 0
  Monocytes-WITHIN-BELOW: number analyzed (Participants) | 97 | 95 | 96 | 98 | 99 | 96 | 98 | 94 | 97 | 98
  Monocytes-WITHIN-BELOW | 5 | 0 | 2 | 0 | 1 | 3 | 2 | 1 | 4 | 3
  Monocytes-WITHIN-WITHIN: number analyzed (Participants) | 97 | 95 | 96 | 98 | 99 | 96 | 98 | 94 | 97 | 98
  Monocytes-WITHIN-WITHIN | 91 | 94 | 94 | 97 | 92 | 91 | 96 | 92 | 93 | 95
  Monocytes-WITHIN-ABOVE: number analyzed (Participants) | 97 | 95 | 96 | 98 | 99 | 96 | 98 | 94 | 97 | 98
  Monocytes-WITHIN-ABOVE | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
  Neutrophils-BELOW-BELOW: number analyzed (Participants) | 1 | 1 | 3 | 4 | 1 | 4 | 3 | 1 | 2 | 7
  Neutrophils-BELOW-BELOW | 1 | 0 | 2 | 1 | 1 | 1 | 2 | 0 | 1 | 5
  Neutrophils-BELOW-WITHIN: number analyzed (Participants) | 1 | 1 | 3 | 4 | 1 | 4 | 3 | 1 | 2 | 7
  Neutrophils-BELOW-WITHIN | 0 | 1 | 1 | 3 | 0 | 3 | 1 | 1 | 1 | 2
  Neutrophils-WITHIN-UNKNOWN: number analyzed (Participants) | 100 | 96 | 96 | 93 | 99 | 94 | 98 | 98 | 99 | 93
  Neutrophils-WITHIN-UNKNOWN | 0 | 1 | 0 | 1 | 4 | 2 | 0 | 0 | 0 | 0
  Neutrophils-WITHIN-BELOW: number analyzed (Participants) | 100 | 96 | 96 | 93 | 99 | 94 | 98 | 98 | 99 | 93
  Neutrophils-WITHIN-BELOW | 2 | 1 | 1 | 2 | 2 | 2 | 0 | 1 | 1 | 0
  Neutrophils-WITHIN-WITHIN: number analyzed (Participants) | 100 | 96 | 96 | 93 | 99 | 94 | 98 | 98 | 99 | 93
  Neutrophils-WITHIN-WITHIN | 98 | 94 | 95 | 89 | 92 | 88 | 98 | 96 | 96 | 93
  Neutrophils-WITHIN-ABOVE: number analyzed (Participants) | 100 | 96 | 96 | 93 | 99 | 94 | 98 | 98 | 99 | 93
  Neutrophils-WITHIN-ABOVE | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 2 | 0
  Neutrophils-ABOVE-WITHIN: number analyzed (Participants) | 0 | 0 | 0 | 3 | 0 | 2 | 2 | 1 | 0 | 1
  Neutrophils-ABOVE-WITHIN | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 1 | 0 | 1
  Neutrophils-ABOVE-ABOVE: number analyzed (Participants) | 0 | 0 | 0 | 3 | 0 | 2 | 2 | 1 | 0 | 1
  Neutrophils-ABOVE-ABOVE | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets-UNKNOWN-UNKNOWN: number analyzed (Participants) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets-UNKNOWN-UNKNOWN | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets-BELOW-BELOW: number analyzed (Participants) | 3 | 1 | 3 | 1 | 2 | 3 | 2 | 1 | 2 | 2
  Platelets-BELOW-BELOW | 3 | 1 | 2 | 1 | 1 | 2 | 0 | 1 | 1 | 2
  Platelets-BELOW-WITHIN: number analyzed (Participants) | 3 | 1 | 3 | 1 | 2 | 3 | 2 | 1 | 2 | 2
  Platelets-BELOW-WITHIN | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0
  Platelets-WITHIN-UNKNOWN: number analyzed (Participants) | 97 | 96 | 95 | 97 | 98 | 96 | 101 | 97 | 98 | 96
  Platelets-WITHIN-UNKNOWN | 1 | 1 | 0 | 3 | 6 | 3 | 2 | 0 | 1 | 0
  Platelets-WITHIN-BELOW: number analyzed (Participants) | 97 | 96 | 95 | 97 | 98 | 96 | 101 | 97 | 98 | 96
  Platelets-WITHIN-BELOW | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
  Platelets-WITHIN-WITHIN: number analyzed (Participants) | 97 | 96 | 95 | 97 | 98 | 96 | 101 | 97 | 98 | 96
  Platelets-WITHIN-WITHIN | 96 | 94 | 94 | 93 | 90 | 93 | 97 | 96 | 96 | 96
  Platelets-WITHIN-ABOVE: number analyzed (Participants) | 97 | 96 | 95 | 97 | 98 | 96 | 101 | 97 | 98 | 96
  Platelets-WITHIN-ABOVE | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0
  Platelets-ABOVE-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 3
  Platelets-ABOVE-WITHIN | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Platelets-ABOVE-ABOVE: number analyzed (Participants) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 3
  Platelets-ABOVE-ABOVE | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 3
  Urea Nitrogen-BELOW-BELOW: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Urea Nitrogen-BELOW-BELOW | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Urea Nitrogen-WITHIN-UNKNOWN: number analyzed (Participants) | 98 | 97 | 98 | 98 | 98 | 93 | 99 | 98 | 100 | 100
  Urea Nitrogen-WITHIN-UNKNOWN | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  Urea Nitrogen-WITHIN-BELOW: number analyzed (Participants) | 98 | 97 | 98 | 98 | 98 | 93 | 99 | 98 | 100 | 100
  Urea Nitrogen-WITHIN-BELOW | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Urea Nitrogen-WITHIN-WITHIN: number analyzed (Participants) | 98 | 97 | 98 | 98 | 98 | 93 | 99 | 98 | 100 | 100
  Urea Nitrogen-WITHIN-WITHIN | 97 | 96 | 95 | 95 | 97 | 93 | 96 | 96 | 98 | 98
  Urea Nitrogen-WITHIN-ABOVE: number analyzed (Participants) | 98 | 97 | 98 | 98 | 98 | 93 | 99 | 98 | 100 | 100
  Urea Nitrogen-WITHIN-ABOVE | 1 | 1 | 3 | 2 | 1 | 0 | 2 | 2 | 1 | 1
  Urea Nitrogen-ABOVE-WITHIN: number analyzed (Participants) | 3 | 0 | 1 | 1 | 2 | 7 | 3 | 2 | 1 | 1
  Urea Nitrogen-ABOVE-WITHIN | 0 | 0 | 1 | 0 | 2 | 5 | 2 | 2 | 0 | 1
  Urea Nitrogen-ABOVE-ABOVE: number analyzed (Participants) | 3 | 0 | 1 | 1 | 2 | 7 | 3 | 2 | 1 | 1
  Urea Nitrogen-ABOVE-ABOVE | 3 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 1 | 0
  Uric Acid-BELOW-BELOW: number analyzed (Participants) | 1 | 2 | 0 | 3 | 0 | 2 | 7 | 4 | 2 | 3
  Uric Acid-BELOW-BELOW | 1 | 0 | 0 | 3 | 0 | 1 | 5 | 3 | 2 | 2
  Uric Acid-BELOW-WITHIN: number analyzed (Participants) | 1 | 2 | 0 | 3 | 0 | 2 | 7 | 4 | 2 | 3
  Uric Acid-BELOW-WITHIN | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1
  Uric Acid-WITHIN-UNKNOWN: number analyzed (Participants) | 95 | 94 | 96 | 96 | 99 | 93 | 93 | 91 | 96 | 94
  Uric Acid-WITHIN-UNKNOWN | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
  Uric Acid-WITHIN-BELOW: number analyzed (Participants) | 95 | 94 | 96 | 96 | 99 | 93 | 93 | 91 | 96 | 94
  Uric Acid-WITHIN-BELOW | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 0 | 1
  Uric Acid-WITHIN-WITHIN: number analyzed (Participants) | 95 | 94 | 96 | 96 | 99 | 93 | 93 | 91 | 96 | 94
  Uric Acid-WITHIN-WITHIN | 94 | 91 | 96 | 93 | 98 | 90 | 89 | 88 | 95 | 89
  Uric Acid-WITHIN-ABOVE: number analyzed (Participants) | 95 | 94 | 96 | 96 | 99 | 93 | 93 | 91 | 96 | 94
  Uric Acid-WITHIN-ABOVE | 1 | 3 | 0 | 2 | 1 | 1 | 3 | 1 | 0 | 3
  Uric Acid-ABOVE-WITHIN: number analyzed (Participants) | 5 | 1 | 3 | 1 | 1 | 5 | 3 | 5 | 3 | 4
  Uric Acid-ABOVE-WITHIN | 2 | 1 | 1 | 0 | 1 | 2 | 2 | 2 | 3 | 2
  Uric Acid-ABOVE-ABOVE: number analyzed (Participants) | 5 | 1 | 3 | 1 | 1 | 5 | 3 | 5 | 3 | 4
  Uric Acid-ABOVE-ABOVE | 3 | 0 | 2 | 1 | 0 | 3 | 1 | 3 | 0 | 2
  White Blood Cells-BELOW-UNKNOWN: number analyzed (Participants) | 3 | 1 | 4 | 6 | 3 | 5 | 5 | 4 | 5 | 10
  White Blood Cells-BELOW-UNKNOWN | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  White Blood Cells-BELOW-BELOW: number analyzed (Participants) | 3 | 1 | 4 | 6 | 3 | 5 | 5 | 4 | 5 | 10
  White Blood Cells-BELOW-BELOW | 1 | 0 | 2 | 2 | 2 | 1 | 3 | 0 | 1 | 4
  White Blood Cells-BELOW-WITHIN: number analyzed (Participants) | 3 | 1 | 4 | 6 | 3 | 5 | 5 | 4 | 5 | 10
  White Blood Cells-BELOW-WITHIN | 2 | 1 | 2 | 4 | 1 | 3 | 2 | 4 | 4 | 6
  White Blood Cells-WITHIN-UNKNOWN: number analyzed (Participants) | 96 | 95 | 95 | 91 | 95 | 93 | 96 | 94 | 95 | 91
  White Blood Cells-WITHIN-UNKNOWN | 0 | 1 | 0 | 1 | 4 | 1 | 0 | 0 | 0 | 0
  White Blood Cells-WITHIN-BELOW: number analyzed (Participants) | 96 | 95 | 95 | 91 | 95 | 93 | 96 | 94 | 95 | 91
  White Blood Cells-WITHIN-BELOW | 2 | 2 | 3 | 2 | 1 | 3 | 1 | 1 | 0 | 1
  White Blood Cells-WITHIN-WITHIN: number analyzed (Participants) | 96 | 95 | 95 | 91 | 95 | 93 | 96 | 94 | 95 | 91
  White Blood Cells-WITHIN-WITHIN | 94 | 91 | 91 | 87 | 89 | 87 | 95 | 91 | 93 | 90
  White Blood Cells-WITHIN-ABOVE: number analyzed (Participants) | 96 | 95 | 95 | 91 | 95 | 93 | 96 | 94 | 95 | 91
  White Blood Cells-WITHIN-ABOVE | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 2 | 2 | 0
  White Blood Cells-ABOVE-WITHIN: number analyzed (Participants) | 2 | 1 | 0 | 3 | 2 | 2 | 2 | 2 | 1 | 0
  White Blood Cells-ABOVE-WITHIN | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 1 | 0
  White Blood Cells-ABOVE-ABOVE: number analyzed (Participants) | 2 | 1 | 0 | 3 | 2 | 2 | 2 | 2 | 1 | 0
  White Blood Cells-ABOVE-ABOVE | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0

8. Primary Outcome: Number of Subjects Presenting Change From Baseline in Hematology and Biochemistry With Respect of Normal Laboratory Ranges, After Second Vaccine Dose (Part A Groups)
Description: Assessed hematological laboratory parameters include basophils, eosinophils, erythrocytes, hemoglobin, lymphocytes, monocytes, neutrophils, platelets, white blood cells. Biochemical laboratory parameters include alanine aminotransferase [ALT], aspartate aminotransferase [AST], creatinine, urea nitrogen and uric acid. Categories reported when comparing Day 61 (pre-vaccination dose 2=baseline) and Day 68 hematological and biochemical laboratory results are defined as follows: <parameter>-<range at baseline>-<range at timing> (e.g. ALT-Within-Within). Ranges level being classified as unknown, below, within or above the normal ranges.
Time Frame: At baseline and at 7 days after the second vaccine dose (Day 68)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group
Number analyzed (Participants) | 12 | 10 | 11 | 12
Participants
  ALT-WITHIN-WITHIN: number analyzed (Participants) | 12 | 10 | 10 | 12
  ALT-WITHIN-WITHIN | 11 | 10 | 10 | 12
  ALT-WITHIN-ABOVE: number analyzed (Participants) | 12 | 10 | 10 | 12
  ALT-WITHIN-ABOVE | 1 | 0 | 0 | 0
  ALT-ABOVE-WITHIN: number analyzed (Participants) | 0 | 0 | 1 | 0
  ALT-ABOVE-WITHIN | 0 | 0 | 1 | 0
  AST-WITHIN-WITHIN: number analyzed (Participants) | 11 | 10 | 11 | 12
  AST-WITHIN-WITHIN | 10 | 10 | 11 | 12
  AST-WITHIN-ABOVE: number analyzed (Participants) | 11 | 10 | 11 | 12
  AST-WITHIN-ABOVE | 1 | 0 | 0 | 0
  AST-ABOVE-ABOVE: number analyzed (Participants) | 1 | 0 | 0 | 0
  AST-ABOVE-ABOVE | 1 | 0 | 0 | 0
  Basophils-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 0
  Basophils-UNKNOWN-WITHIN | 1 | 0 | 0 | 0
  Basophils-WITHIN-WITHIN: number analyzed (Participants) | 11 | 10 | 11 | 12
  Basophils-WITHIN-WITHIN | 11 | 10 | 11 | 12
  Creatinine-BELOW-BELOW: number analyzed (Participants) | 0 | 0 | 0 | 1
  Creatinine-BELOW-BELOW | 0 | 0 | 0 | 1
  Creatinine-WITHIN-WITHIN: number analyzed (Participants) | 12 | 9 | 11 | 10
  Creatinine-WITHIN-WITHIN | 12 | 7 | 11 | 10
  Creatinine-WITHIN-ABOVE: number analyzed (Participants) | 12 | 9 | 11 | 10
  Creatinine-WITHIN-ABOVE | 0 | 2 | 0 | 0
  Creatinine-ABOVE-WITHIN: number analyzed (Participants) | 0 | 1 | 0 | 1
  Creatinine-ABOVE-WITHIN | 0 | 0 | 0 | 1
  Creatinine-ABOVE-ABOVE: number analyzed (Participants) | 0 | 1 | 0 | 1
  Creatinine-ABOVE-ABOVE | 0 | 1 | 0 | 0
  Eosinophils-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 0
  Eosinophils-UNKNOWN-WITHIN | 1 | 0 | 0 | 0
  Eosinophils-BELOW-BELOW: number analyzed (Participants) | 0 | 1 | 1 | 0
  Eosinophils-BELOW-BELOW | 0 | 0 | 1 | 0
  Eosinophils-BELOW-WITHIN: number analyzed (Participants) | 0 | 1 | 1 | 0
  Eosinophils-BELOW-WITHIN | 0 | 1 | 0 | 0
  Eosinophils-WITHIN-BELOW: number analyzed (Participants) | 11 | 9 | 10 | 12
  Eosinophils-WITHIN-BELOW | 1 | 0 | 1 | 0
  Eosinophils-WITHIN-WITHIN: number analyzed (Participants) | 11 | 9 | 10 | 12
  Eosinophils-WITHIN-WITHIN | 10 | 9 | 8 | 12
  Eosinophils-WITHIN-ABOVE: number analyzed (Participants) | 11 | 9 | 10 | 12
  Eosinophils-WITHIN-ABOVE | 0 | 0 | 1 | 0
  Erythrocytes-UNKNOWN-BELOW: number analyzed (Participants) | 1 | 0 | 0 | 0
  Erythrocytes-UNKNOWN-BELOW | 1 | 0 | 0 | 0
  Erythrocytes-WITHIN-BELOW: number analyzed (Participants) | 11 | 9 | 11 | 12
  Erythrocytes-WITHIN-BELOW | 1 | 0 | 0 | 0
  Erythrocytes-WITHIN-WITHIN: number analyzed (Participants) | 11 | 9 | 11 | 12
  Erythrocytes-WITHIN-WITHIN | 10 | 9 | 10 | 12
  Erythrocytes-WITHIN-ABOVE: number analyzed (Participants) | 11 | 9 | 11 | 12
  Erythrocytes-WITHIN-ABOVE | 0 | 0 | 1 | 0
  Erythrocytes-ABOVE-ABOVE: number analyzed (Participants) | 0 | 1 | 0 | 0
  Erythrocytes-ABOVE-ABOVE | 0 | 1 | 0 | 0
  Hemoglobin-UNKNOWN-BELOW: number analyzed (Participants) | 1 | 0 | 0 | 0
  Hemoglobin-UNKNOWN-BELOW | 1 | 0 | 0 | 0
  Hemoglobin-BELOW-WITHIN: number analyzed (Participants) | 0 | 0 | 1 | 0
  Hemoglobin-BELOW-WITHIN | 0 | 0 | 1 | 0
  Hemoglobin-WITHIN-WITHIN: number analyzed (Participants) | 11 | 10 | 10 | 12
  Hemoglobin-WITHIN-WITHIN | 11 | 10 | 9 | 12
  Hemoglobin-WITHIN-ABOVE: number analyzed (Participants) | 11 | 10 | 10 | 12
  Hemoglobin-WITHIN-ABOVE | 0 | 0 | 1 | 0
  Lymphocytes-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 0
  Lymphocytes-UNKNOWN-WITHIN | 1 | 0 | 0 | 0
  Lymphocytes-BELOW-WITHIN: number analyzed (Participants) | 0 | 0 | 0 | 1
  Lymphocytes-BELOW-WITHIN | 0 | 0 | 0 | 1
  Lymphocytes-WITHIN-WITHIN: number analyzed (Participants) | 11 | 10 | 11 | 11
  Lymphocytes-WITHIN-WITHIN | 11 | 10 | 11 | 11
  Monocytes-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 0
  Monocytes-UNKNOWN-WITHIN | 1 | 0 | 0 | 0
  Monocytes-BELOW-WITHIN: number analyzed (Participants) | 0 | 0 | 1 | 0
  Monocytes-BELOW-WITHIN | 0 | 0 | 1 | 0
  Monocytes-WITHIN-WITHIN: number analyzed (Participants) | 11 | 10 | 10 | 12
  Monocytes-WITHIN-WITHIN | 11 | 10 | 10 | 12
  Neutrophils-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 0
  Neutrophils-UNKNOWN-WITHIN | 1 | 0 | 0 | 0
  Neutrophils-BELOW-BELOW: number analyzed (Participants) | 1 | 0 | 1 | 0
  Neutrophils-BELOW-BELOW | 0 | 0 | 1 | 0
  Neutrophils-BELOW-WITHIN: number analyzed (Participants) | 1 | 0 | 1 | 0
  Neutrophils-BELOW-WITHIN | 1 | 0 | 0 | 0
  Neutrophils-WITHIN-BELOW: number analyzed (Participants) | 10 | 10 | 10 | 12
  Neutrophils-WITHIN-BELOW | 1 | 0 | 0 | 0
  Neutrophils-WITHIN-WITHIN: number analyzed (Participants) | 10 | 10 | 10 | 12
  Neutrophils-WITHIN-WITHIN | 9 | 10 | 10 | 12
  Platelets-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 1 | 0 | 0
  Platelets-UNKNOWN-WITHIN | 1 | 1 | 0 | 0
  Platelets-WITHIN-WITHIN: number analyzed (Participants) | 11 | 8 | 11 | 12
  Platelets-WITHIN-WITHIN | 11 | 8 | 11 | 12
  Platelets-ABOVE-WITHIN: number analyzed (Participants) | 0 | 1 | 0 | 0
  Platelets-ABOVE-WITHIN | 0 | 1 | 0 | 0
  Urea Nitrogen-WITHIN-WITHIN | 12 | 10 | 11 | 12
  Uric Acid-BELOW-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 0
  Uric Acid-BELOW-WITHIN | 1 | 0 | 0 | 0
  Uric Acid-WITHIN-WITHIN: number analyzed (Participants) | 11 | 10 | 11 | 12
  Uric Acid-WITHIN-WITHIN | 11 | 10 | 11 | 12
  White Blood Cells-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 0
  White Blood Cells-UNKNOWN-WITHIN | 1 | 0 | 0 | 0
  White Blood Cells-BELOW-BELOW: number analyzed (Participants) | 2 | 0 | 1 | 0
  White Blood Cells-BELOW-BELOW | 1 | 0 | 1 | 0
  White Blood Cells-BELOW-WITHIN: number analyzed (Participants) | 2 | 0 | 1 | 0
  White Blood Cells-BELOW-WITHIN | 1 | 0 | 0 | 0
  White Blood Cells-WITHIN-BELOW: number analyzed (Participants) | 8 | 10 | 10 | 12
  White Blood Cells-WITHIN-BELOW | 1 | 0 | 0 | 0
  White Blood Cells-WITHIN-WITHIN: number analyzed (Participants) | 8 | 10 | 10 | 12
  White Blood Cells-WITHIN-WITHIN | 7 | 10 | 10 | 12
  White Blood Cells-ABOVE-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 0
  White Blood Cells-ABOVE-WITHIN | 1 | 0 | 0 | 0

9. Primary Outcome: Number of Subjects Presenting Change From Baseline in Hematology and Biochemistry With Respect of Normal Laboratory Ranges, After Second Vaccine Dose (Part B Groups)
Description: as for outcome 8
Time Frame: At baseline and at 7 days after the second vaccine dose (Day 68)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 97 | 94 | 95 | 96 | 98 | 97 | 98 | 97 | 97 | 99
Participants
  ALT-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0
  ALT-UNKNOWN-WITHIN | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0
  ALT-WITHIN-UNKNOWN: number analyzed (Participants) | 95 | 94 | 95 | 93 | 96 | 96 | 95 | 93 | 91 | 97
  ALT-WITHIN-UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  ALT-WITHIN-WITHIN: number analyzed (Participants) | 95 | 94 | 95 | 93 | 96 | 96 | 95 | 93 | 91 | 97
  ALT-WITHIN-WITHIN | 93 | 94 | 95 | 93 | 94 | 94 | 95 | 91 | 90 | 96
  ALT-WITHIN-ABOVE: number analyzed (Participants) | 95 | 94 | 95 | 93 | 96 | 96 | 95 | 93 | 91 | 97
  ALT-WITHIN-ABOVE | 2 | 0 | 0 | 0 | 2 | 2 | 0 | 2 | 1 | 0
  ALT-ABOVE-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 2 | 2 | 0 | 2 | 3 | 4 | 2
  ALT-ABOVE-WITHIN | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 2 | 0
  ALT-ABOVE-ABOVE: number analyzed (Participants) | 1 | 0 | 0 | 2 | 2 | 0 | 2 | 3 | 4 | 2
  ALT-ABOVE-ABOVE | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 2
  AST-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0
  AST-UNKNOWN-WITHIN | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0
  AST-WITHIN-UNKNOWN: number analyzed (Participants) | 96 | 93 | 95 | 94 | 97 | 96 | 95 | 95 | 93 | 98
  AST-WITHIN-UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  AST-WITHIN-WITHIN: number analyzed (Participants) | 96 | 93 | 95 | 94 | 97 | 96 | 95 | 95 | 93 | 98
  AST-WITHIN-WITHIN | 94 | 93 | 95 | 93 | 97 | 94 | 95 | 93 | 92 | 97
  AST-WITHIN-ABOVE: number analyzed (Participants) | 96 | 93 | 95 | 94 | 97 | 96 | 95 | 95 | 93 | 98
  AST-WITHIN-ABOVE | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 1 | 0
  AST-ABOVE-WITHIN: number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 1
  AST-ABOVE-WITHIN | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
  AST-ABOVE-ABOVE: number analyzed (Participants) | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 1
  AST-ABOVE-ABOVE | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 1
  Basophils-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Basophils-UNKNOWN-WITHIN | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Basophils-WITHIN-UNKNOWN: number analyzed (Participants) | 96 | 94 | 94 | 96 | 96 | 95 | 96 | 96 | 95 | 98
  Basophils-WITHIN-UNKNOWN | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Basophils-WITHIN-WITHIN: number analyzed (Participants) | 96 | 94 | 94 | 96 | 96 | 95 | 96 | 96 | 95 | 98
  Basophils-WITHIN-WITHIN | 95 | 94 | 94 | 96 | 95 | 94 | 96 | 96 | 95 | 97
  Creatinine-UNKNOWN-BELOW: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0
  Creatinine-UNKNOWN-BELOW | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0
  Creatinine-UNKNOWN-WITHIN | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
  Creatinine-UNKNOWN-ABOVE: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0
  Creatinine-UNKNOWN-ABOVE | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Creatinine-BELOW-UNKNOWN: number analyzed (Participants) | 3 | 6 | 3 | 3 | 4 | 1 | 3 | 6 | 7 | 1
  Creatinine-BELOW-UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Creatinine-BELOW-BELOW: number analyzed (Participants) | 3 | 6 | 3 | 3 | 4 | 1 | 3 | 6 | 7 | 1
  Creatinine-BELOW-BELOW | 0 | 4 | 2 | 2 | 4 | 1 | 2 | 3 | 1 | 0
  Creatinine-BELOW-WITHIN: number analyzed (Participants) | 3 | 6 | 3 | 3 | 4 | 1 | 3 | 6 | 7 | 1
  Creatinine-BELOW-WITHIN | 3 | 2 | 1 | 1 | 0 | 0 | 1 | 3 | 6 | 0
  Creatinine-WITHIN-BELOW: number analyzed (Participants) | 87 | 83 | 90 | 89 | 92 | 94 | 93 | 88 | 87 | 97
  Creatinine-WITHIN-BELOW | 1 | 2 | 2 | 2 | 3 | 3 | 2 | 1 | 1 | 0
  Creatinine-WITHIN-WITHIN: number analyzed (Participants) | 87 | 83 | 90 | 89 | 92 | 94 | 93 | 88 | 87 | 97
  Creatinine-WITHIN-WITHIN | 83 | 81 | 86 | 87 | 88 | 90 | 88 | 86 | 83 | 96
  Creatinine-WITHIN-ABOVE: number analyzed (Participants) | 87 | 83 | 90 | 89 | 92 | 94 | 93 | 88 | 87 | 97
  Creatinine-WITHIN-ABOVE | 3 | 0 | 2 | 0 | 1 | 1 | 3 | 1 | 3 | 1
  Creatinine-ABOVE-WITHIN: number analyzed (Participants) | 6 | 5 | 2 | 3 | 2 | 1 | 1 | 2 | 1 | 1
  Creatinine-ABOVE-WITHIN | 2 | 2 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0
  Creatinine-ABOVE-ABOVE: number analyzed (Participants) | 6 | 5 | 2 | 3 | 2 | 1 | 1 | 2 | 1 | 1
  Creatinine-ABOVE-ABOVE | 4 | 3 | 2 | 1 | 1 | 1 | 0 | 2 | 1 | 1
  Eosinophils-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Eosinophils-UNKNOWN-WITHIN | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 2 | 1
  Eosinophils-UNKNOWN-ABOVE: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Eosinophils-UNKNOWN-ABOVE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Eosinophils-BELOW-UNKNOWN: number analyzed (Participants) | 7 | 5 | 9 | 6 | 8 | 5 | 6 | 8 | 6 | 8
  Eosinophils-BELOW-UNKNOWN | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Eosinophils-BELOW-BELOW: number analyzed (Participants) | 7 | 5 | 9 | 6 | 8 | 5 | 6 | 8 | 6 | 8
  Eosinophils-BELOW-BELOW | 3 | 2 | 4 | 2 | 3 | 4 | 1 | 1 | 4 | 3
  Eosinophils-BELOW-WITHIN: number analyzed (Participants) | 7 | 5 | 9 | 6 | 8 | 5 | 6 | 8 | 6 | 8
  Eosinophils-BELOW-WITHIN | 3 | 3 | 5 | 4 | 5 | 1 | 5 | 7 | 2 | 5
  Eosinophils-WITHIN-UNKNOWN: number analyzed (Participants) | 86 | 87 | 82 | 87 | 84 | 88 | 85 | 87 | 87 | 88
  Eosinophils-WITHIN-UNKNOWN | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Eosinophils-WITHIN-BELOW: number analyzed (Participants) | 86 | 87 | 82 | 87 | 84 | 88 | 85 | 87 | 87 | 88
  Eosinophils-WITHIN-BELOW | 2 | 2 | 4 | 6 | 3 | 1 | 6 | 1 | 3 | 0
  Eosinophils-WITHIN-WITHIN: number analyzed (Participants) | 86 | 87 | 82 | 87 | 84 | 88 | 85 | 87 | 87 | 88
  Eosinophils-WITHIN-WITHIN | 82 | 85 | 78 | 79 | 79 | 83 | 78 | 83 | 83 | 87
  Eosinophils-WITHIN-ABOVE: number analyzed (Participants) | 86 | 87 | 82 | 87 | 84 | 88 | 85 | 87 | 87 | 88
  Eosinophils-WITHIN-ABOVE | 2 | 0 | 0 | 2 | 1 | 3 | 1 | 3 | 1 | 0
  Eosinophils-ABOVE-WITHIN: number analyzed (Participants) | 3 | 2 | 3 | 3 | 4 | 2 | 5 | 1 | 2 | 2
  Eosinophils-ABOVE-WITHIN | 1 | 1 | 2 | 2 | 0 | 1 | 4 | 1 | 0 | 2
  Eosinophils-ABOVE-ABOVE: number analyzed (Participants) | 3 | 2 | 3 | 3 | 4 | 2 | 5 | 1 | 2 | 2
  Eosinophils-ABOVE-ABOVE | 2 | 1 | 1 | 1 | 4 | 1 | 1 | 0 | 2 | 0
  Erythrocytes-UNKNOWN-BELOW: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Erythrocytes-UNKNOWN-BELOW | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Erythrocytes-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Erythrocytes-UNKNOWN-WITHIN | 1 | 0 | 1 | 0 | 1 | 2 | 2 | 1 | 2 | 0
  Erythrocytes-UNKNOWN-ABOVE: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Erythrocytes-UNKNOWN-ABOVE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Erythrocytes-BELOW-BELOW: number analyzed (Participants) | 7 | 2 | 0 | 2 | 3 | 4 | 3 | 0 | 4 | 1
  Erythrocytes-BELOW-BELOW | 6 | 2 | 0 | 1 | 3 | 4 | 2 | 0 | 2 | 1
  Erythrocytes-BELOW-WITHIN: number analyzed (Participants) | 7 | 2 | 0 | 2 | 3 | 4 | 3 | 0 | 4 | 1
  Erythrocytes-BELOW-WITHIN | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0
  Erythrocytes-WITHIN-UNKNOWN: number analyzed (Participants) | 87 | 91 | 91 | 93 | 92 | 89 | 90 | 94 | 90 | 96
  Erythrocytes-WITHIN-UNKNOWN | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Erythrocytes-WITHIN-BELOW: number analyzed (Participants) | 87 | 91 | 91 | 93 | 92 | 89 | 90 | 94 | 90 | 96
  Erythrocytes-WITHIN-BELOW | 3 | 3 | 0 | 1 | 2 | 3 | 1 | 0 | 1 | 3
  Erythrocytes-WITHIN-WITHIN: number analyzed (Participants) | 87 | 91 | 91 | 93 | 92 | 89 | 90 | 94 | 90 | 96
  Erythrocytes-WITHIN-WITHIN | 83 | 88 | 91 | 92 | 89 | 83 | 89 | 94 | 89 | 92
  Erythrocytes-WITHIN-ABOVE: number analyzed (Participants) | 87 | 91 | 91 | 93 | 92 | 89 | 90 | 94 | 90 | 96
  Erythrocytes-WITHIN-ABOVE | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Erythrocytes-ABOVE-WITHIN: number analyzed (Participants) | 2 | 1 | 3 | 1 | 1 | 2 | 3 | 2 | 1 | 1
  Erythrocytes-ABOVE-WITHIN | 2 | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 0
  Erythrocytes-ABOVE-ABOVE: number analyzed (Participants) | 2 | 1 | 3 | 1 | 1 | 2 | 3 | 2 | 1 | 1
  Erythrocytes-ABOVE-ABOVE | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 2 | 1 | 1
  Hemoglobin-UNKNOWN-BELOW: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Hemoglobin-UNKNOWN-BELOW | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Hemoglobin-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Hemoglobin-UNKNOWN-WITHIN | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 2 | 1
  Hemoglobin-BELOW-BELOW: number analyzed (Participants) | 8 | 8 | 3 | 7 | 5 | 9 | 6 | 3 | 9 | 4
  Hemoglobin-BELOW-BELOW | 7 | 6 | 2 | 6 | 3 | 6 | 5 | 3 | 8 | 3
  Hemoglobin-BELOW-WITHIN: number analyzed (Participants) | 8 | 8 | 3 | 7 | 5 | 9 | 6 | 3 | 9 | 4
  Hemoglobin-BELOW-WITHIN | 1 | 2 | 1 | 1 | 2 | 3 | 1 | 0 | 1 | 1
  Hemoglobin-WITHIN-UNKNOWN: number analyzed (Participants) | 87 | 85 | 90 | 86 | 90 | 84 | 90 | 91 | 85 | 94
  Hemoglobin-WITHIN-UNKNOWN | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Hemoglobin-WITHIN-BELOW: number analyzed (Participants) | 87 | 85 | 90 | 86 | 90 | 84 | 90 | 91 | 85 | 94
  Hemoglobin-WITHIN-BELOW | 5 | 2 | 0 | 0 | 3 | 1 | 1 | 1 | 3 | 2
  Hemoglobin-WITHIN-WITHIN: number analyzed (Participants) | 87 | 85 | 90 | 86 | 90 | 84 | 90 | 91 | 85 | 94
  Hemoglobin-WITHIN-WITHIN | 81 | 83 | 89 | 86 | 86 | 82 | 89 | 90 | 82 | 91
  Hemoglobin-WITHIN-ABOVE: number analyzed (Participants) | 87 | 85 | 90 | 86 | 90 | 84 | 90 | 91 | 85 | 94
  Hemoglobin-WITHIN-ABOVE | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin-ABOVE-WITHIN: number analyzed (Participants) | 1 | 1 | 1 | 3 | 1 | 2 | 0 | 2 | 1 | 0
  Hemoglobin-ABOVE-WITHIN | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 1 | 0 | 0
  Hemoglobin-ABOVE-ABOVE: number analyzed (Participants) | 1 | 1 | 1 | 3 | 1 | 2 | 0 | 2 | 1 | 0
  Hemoglobin-ABOVE-ABOVE | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0
  Lymphocytes-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Lymphocytes-UNKNOWN-WITHIN | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Lymphocytes-BELOW-BELOW: number analyzed (Participants) | 2 | 1 | 4 | 4 | 4 | 2 | 3 | 1 | 1 | 5
  Lymphocytes-BELOW-BELOW | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 0 | 4
  Lymphocytes-BELOW-WITHIN: number analyzed (Participants) | 2 | 1 | 4 | 4 | 4 | 2 | 3 | 1 | 1 | 5
  Lymphocytes-BELOW-WITHIN | 2 | 1 | 4 | 2 | 3 | 1 | 1 | 1 | 1 | 1
  Lymphocytes-WITHIN-UNKNOWN: number analyzed (Participants) | 93 | 92 | 90 | 91 | 91 | 93 | 93 | 95 | 94 | 93
  Lymphocytes-WITHIN-UNKNOWN | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Lymphocytes-WITHIN-BELOW: number analyzed (Participants) | 93 | 92 | 90 | 91 | 91 | 93 | 93 | 95 | 94 | 93
  Lymphocytes-WITHIN-BELOW | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 0 | 1
  Lymphocytes-WITHIN-WITHIN: number analyzed (Participants) | 93 | 92 | 90 | 91 | 91 | 93 | 93 | 95 | 94 | 93
  Lymphocytes-WITHIN-WITHIN | 90 | 91 | 89 | 90 | 88 | 92 | 91 | 94 | 94 | 91
  Lymphocytes-WITHIN-ABOVE: number analyzed (Participants) | 93 | 92 | 90 | 91 | 91 | 93 | 93 | 95 | 94 | 93
  Lymphocytes-WITHIN-ABOVE | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocytes-ABOVE-WITHIN: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocytes-ABOVE-WITHIN | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes-ABOVE-ABOVE: number analyzed (Participants) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Lymphocytes-ABOVE-ABOVE | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Monocytes-UNKNOWN-BELOW: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Monocytes-UNKNOWN-BELOW | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Monocytes-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Monocytes-UNKNOWN-WITHIN | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 1 | 1
  Monocytes-BELOW-BELOW: number analyzed (Participants) | 5 | 0 | 4 | 3 | 4 | 6 | 4 | 4 | 5 | 6
  Monocytes-BELOW-BELOW | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 3
  Monocytes-BELOW-WITHIN: number analyzed (Participants) | 5 | 0 | 4 | 3 | 4 | 6 | 4 | 4 | 5 | 6
  Monocytes-BELOW-WITHIN | 3 | 0 | 4 | 3 | 3 | 5 | 4 | 3 | 4 | 3
  Monocytes-WITHIN-UNKNOWN: number analyzed (Participants) | 89 | 94 | 90 | 93 | 92 | 89 | 92 | 91 | 90 | 92
  Monocytes-WITHIN-UNKNOWN | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Monocytes-WITHIN-BELOW: number analyzed (Participants) | 89 | 94 | 90 | 93 | 92 | 89 | 92 | 91 | 90 | 92
  Monocytes-WITHIN-BELOW | 1 | 2 | 3 | 2 | 1 | 6 | 1 | 3 | 1 | 3
  Monocytes-WITHIN-WITHIN: number analyzed (Participants) | 89 | 94 | 90 | 93 | 92 | 89 | 92 | 91 | 90 | 92
  Monocytes-WITHIN-WITHIN | 87 | 92 | 87 | 91 | 90 | 82 | 91 | 88 | 89 | 88
  Monocytes-ABOVE-WITHIN: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Monocytes-ABOVE-WITHIN | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Monocytes-ABOVE-ABOVE: number analyzed (Participants) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Monocytes-ABOVE-ABOVE | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Neutrophils-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Neutrophils-UNKNOWN-WITHIN | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  Neutrophils-BELOW-BELOW: number analyzed (Participants) | 2 | 1 | 1 | 3 | 1 | 3 | 2 | 1 | 1 | 2
  Neutrophils-BELOW-BELOW | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 2
  Neutrophils-BELOW-WITHIN: number analyzed (Participants) | 2 | 1 | 1 | 3 | 1 | 3 | 2 | 1 | 1 | 2
  Neutrophils-BELOW-WITHIN | 1 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 0
  Neutrophils-WITHIN-UNKNOWN: number analyzed (Participants) | 94 | 92 | 93 | 92 | 95 | 92 | 94 | 95 | 93 | 96
  Neutrophils-WITHIN-UNKNOWN | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  Neutrophils-WITHIN-BELOW: number analyzed (Participants) | 94 | 92 | 93 | 92 | 95 | 92 | 94 | 95 | 93 | 96
  Neutrophils-WITHIN-BELOW | 0 | 1 | 3 | 1 | 1 | 1 | 2 | 0 | 4 | 2
  Neutrophils-WITHIN-WITHIN: number analyzed (Participants) | 94 | 92 | 93 | 92 | 95 | 92 | 94 | 95 | 93 | 96
  Neutrophils-WITHIN-WITHIN | 92 | 90 | 90 | 90 | 91 | 90 | 92 | 95 | 89 | 92
  Neutrophils-WITHIN-ABOVE: number analyzed (Participants) | 94 | 92 | 93 | 92 | 95 | 92 | 94 | 95 | 93 | 96
  Neutrophils-WITHIN-ABOVE | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 1
  Neutrophils-ABOVE-WITHIN: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Neutrophils-ABOVE-WITHIN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Neutrophils-ABOVE-ABOVE: number analyzed (Participants) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Neutrophils-ABOVE-ABOVE | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets-UNKNOWN-UNKNOWN: number analyzed (Participants) | 3 | 2 | 2 | 0 | 2 | 3 | 5 | 2 | 2 | 1
  Platelets-UNKNOWN-UNKNOWN | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Platelets-UNKNOWN-WITHIN: number analyzed (Participants) | 3 | 2 | 2 | 0 | 2 | 3 | 5 | 2 | 2 | 1
  Platelets-UNKNOWN-WITHIN | 2 | 2 | 2 | 0 | 2 | 2 | 5 | 2 | 2 | 1
  Platelets-BELOW-UNKNOWN: number analyzed (Participants) | 3 | 1 | 3 | 1 | 0 | 2 | 1 | 1 | 1 | 2
  Platelets-BELOW-UNKNOWN | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets-BELOW-BELOW: number analyzed (Participants) | 3 | 1 | 3 | 1 | 0 | 2 | 1 | 1 | 1 | 2
  Platelets-BELOW-BELOW | 3 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 2
  Platelets-BELOW-WITHIN: number analyzed (Participants) | 3 | 1 | 3 | 1 | 0 | 2 | 1 | 1 | 1 | 2
  Platelets-BELOW-WITHIN | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  Platelets-WITHIN-UNKNOWN: number analyzed (Participants) | 89 | 91 | 89 | 93 | 96 | 90 | 91 | 92 | 92 | 93
  Platelets-WITHIN-UNKNOWN | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1
  Platelets-WITHIN-BELOW: number analyzed (Participants) | 89 | 91 | 89 | 93 | 96 | 90 | 91 | 92 | 92 | 93
  Platelets-WITHIN-BELOW | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
  Platelets-WITHIN-WITHIN: number analyzed (Participants) | 89 | 91 | 89 | 93 | 96 | 90 | 91 | 92 | 92 | 93
  Platelets-WITHIN-WITHIN | 88 | 89 | 88 | 91 | 92 | 88 | 87 | 90 | 89 | 91
  Platelets-WITHIN-ABOVE: number analyzed (Participants) | 89 | 91 | 89 | 93 | 96 | 90 | 91 | 92 | 92 | 93
  Platelets-WITHIN-ABOVE | 0 | 1 | 1 | 2 | 2 | 0 | 2 | 1 | 3 | 1
  Platelets-ABOVE-WITHIN: number analyzed (Participants) | 2 | 0 | 1 | 2 | 0 | 2 | 1 | 2 | 2 | 3
  Platelets-ABOVE-WITHIN | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  Platelets-ABOVE-ABOVE: number analyzed (Participants) | 2 | 0 | 1 | 2 | 0 | 2 | 1 | 2 | 2 | 3
  Platelets-ABOVE-ABOVE | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 3
  Urea Nitrogen-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0
  Urea Nitrogen-UNKNOWN-WITHIN | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0
  Urea Nitrogen-UNKNOWN-ABOVE: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0
  Urea Nitrogen-UNKNOWN-ABOVE | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Urea Nitrogen-BELOW-BELOW: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0
  Urea Nitrogen-BELOW-BELOW | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  Urea Nitrogen-BELOW-WITHIN: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0
  Urea Nitrogen-BELOW-WITHIN | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
  Urea Nitrogen-WITHIN-UNKNOWN: number analyzed (Participants) | 92 | 94 | 93 | 92 | 95 | 94 | 92 | 92 | 92 | 99
  Urea Nitrogen-WITHIN-UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Urea Nitrogen-WITHIN-WITHIN: number analyzed (Participants) | 92 | 94 | 93 | 92 | 95 | 94 | 92 | 92 | 92 | 99
  Urea Nitrogen-WITHIN-WITHIN | 91 | 94 | 93 | 91 | 95 | 94 | 91 | 91 | 91 | 97
  Urea Nitrogen-WITHIN-ABOVE: number analyzed (Participants) | 92 | 94 | 93 | 92 | 95 | 94 | 92 | 92 | 92 | 99
  Urea Nitrogen-WITHIN-ABOVE | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1
  Urea Nitrogen-ABOVE-WITHIN: number analyzed (Participants) | 4 | 0 | 2 | 2 | 3 | 2 | 3 | 3 | 2 | 0
  Urea Nitrogen-ABOVE-WITHIN | 1 | 0 | 2 | 1 | 3 | 1 | 2 | 2 | 2 | 0
  Urea Nitrogen-ABOVE-ABOVE: number analyzed (Participants) | 4 | 0 | 2 | 2 | 3 | 2 | 3 | 3 | 2 | 0
  Urea Nitrogen-ABOVE-ABOVE | 3 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  Uric Acid-UNKNOWN-BELOW: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0
  Uric Acid-UNKNOWN-BELOW | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Uric Acid-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0
  Uric Acid-UNKNOWN-WITHIN | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
  Uric Acid-UNKNOWN-ABOVE: number analyzed (Participants) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 2 | 0
  Uric Acid-UNKNOWN-ABOVE | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Uric Acid-BELOW-BELOW: number analyzed (Participants) | 2 | 2 | 1 | 3 | 0 | 1 | 4 | 2 | 2 | 3
  Uric Acid-BELOW-BELOW | 1 | 2 | 0 | 3 | 0 | 1 | 4 | 2 | 2 | 2
  Uric Acid-BELOW-WITHIN: number analyzed (Participants) | 2 | 2 | 1 | 3 | 0 | 1 | 4 | 2 | 2 | 3
  Uric Acid-BELOW-WITHIN | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Uric Acid-WITHIN-UNKNOWN: number analyzed (Participants) | 91 | 87 | 92 | 90 | 98 | 92 | 93 | 91 | 92 | 91
  Uric Acid-WITHIN-UNKNOWN | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Uric Acid-WITHIN-BELOW: number analyzed (Participants) | 91 | 87 | 92 | 90 | 98 | 92 | 93 | 91 | 92 | 91
  Uric Acid-WITHIN-BELOW | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 3
  Uric Acid-WITHIN-WITHIN: number analyzed (Participants) | 91 | 87 | 92 | 90 | 98 | 92 | 93 | 91 | 92 | 91
  Uric Acid-WITHIN-WITHIN | 91 | 86 | 87 | 89 | 98 | 91 | 92 | 87 | 91 | 83
  Uric Acid-WITHIN-ABOVE: number analyzed (Participants) | 91 | 87 | 92 | 90 | 98 | 92 | 93 | 91 | 92 | 91
  Uric Acid-WITHIN-ABOVE | 0 | 0 | 4 | 1 | 0 | 0 | 0 | 3 | 1 | 4
  Uric Acid-ABOVE-WITHIN: number analyzed (Participants) | 3 | 5 | 2 | 2 | 0 | 3 | 0 | 3 | 1 | 5
  Uric Acid-ABOVE-WITHIN | 1 | 2 | 1 | 2 | 0 | 2 | 0 | 2 | 1 | 4
  Uric Acid-ABOVE-ABOVE: number analyzed (Participants) | 3 | 5 | 2 | 2 | 0 | 3 | 0 | 3 | 1 | 5
  Uric Acid-ABOVE-ABOVE | 2 | 3 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
  White Blood Cells-UNKNOWN-WITHIN: number analyzed (Participants) | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  White Blood Cells-UNKNOWN-WITHIN | 1 | 0 | 1 | 0 | 2 | 2 | 2 | 1 | 2 | 1
  White Blood Cells-BELOW-BELOW: number analyzed (Participants) | 4 | 0 | 3 | 4 | 5 | 4 | 7 | 4 | 3 | 5
  White Blood Cells-BELOW-BELOW | 2 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 1 | 4
  White Blood Cells-BELOW-WITHIN: number analyzed (Participants) | 4 | 0 | 3 | 4 | 5 | 4 | 7 | 4 | 3 | 5
  White Blood Cells-BELOW-WITHIN | 2 | 0 | 2 | 3 | 4 | 4 | 6 | 2 | 2 | 1
  White Blood Cells-WITHIN-UNKNOWN: number analyzed (Participants) | 91 | 92 | 91 | 90 | 89 | 91 | 89 | 92 | 91 | 93
  White Blood Cells-WITHIN-UNKNOWN | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
  White Blood Cells-WITHIN-BELOW: number analyzed (Participants) | 91 | 92 | 91 | 90 | 89 | 91 | 89 | 92 | 91 | 93
  White Blood Cells-WITHIN-BELOW | 3 | 0 | 2 | 3 | 3 | 2 | 1 | 0 | 3 | 1
  White Blood Cells-WITHIN-WITHIN: number analyzed (Participants) | 91 | 92 | 91 | 90 | 89 | 91 | 89 | 92 | 91 | 93
  White Blood Cells-WITHIN-WITHIN | 86 | 92 | 89 | 86 | 83 | 88 | 88 | 91 | 88 | 90
  White Blood Cells-WITHIN-ABOVE: number analyzed (Participants) | 91 | 92 | 91 | 90 | 89 | 91 | 89 | 92 | 91 | 93
  White Blood Cells-WITHIN-ABOVE | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1
  White Blood Cells-ABOVE-WITHIN: number analyzed (Participants) | 1 | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0
  White Blood Cells-ABOVE-WITHIN | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
  White Blood Cells-ABOVE-ABOVE: number analyzed (Participants) | 1 | 2 | 0 | 2 | 2 | 0 | 0 | 0 | 1 | 0
  White Blood Cells-ABOVE-ABOVE | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Subjects With Any Grade 3 Non-serious AEs (Solicited and Unsolicited) After First Dose of Vaccination
Description: A Grade 3 AE is any AE assessed as severe, i.e. which prevents normal, everyday activities. In adults, such an AE would, for example, prevent attendance at work and would necessitate the administration of corrective therapy.
Time Frame: During a 30-day follow-up period (i.e., on the day of vaccination at Day 1, and 29 subsequent days) after first dose of vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 101 | 97 | 100 | 101 | 101 | 100 | 103 | 100 | 101 | 101
Participants
  Any adverse event | 1 | 0 | 0 | 0 | 1 | 1 | 4 | 3 | 7 | 1 | 7 | 6 | 8 | 4
  General adverse event | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 2 | 5 | 0 | 2 | 3 | 4 | 4
  Local adverse event | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 6 | 3 | 4 | 0

11. Primary Outcome: Number of Subjects With Any Grade 3 Non-serious AEs (Solicited and Unsolicited) After Second Dose of Vaccination
Description: as for outcome 10
Time Frame: During a 30-day follow-up period (i.e., on the day of vaccination at Day 61, and 29 subsequent days) after second dose of vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 12 | 10 | 11 | 12 | 98 | 95 | 95 | 96 | 98 | 97 | 98 | 97 | 97 | 99
Participants
  Any adverse event | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 5 | 3 | 5 | 8 | 7 | 3 | 0
  General adverse event | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 2 | 2 | 5 | 5 | 1 | 0
  Local adverse event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 4 | 2 | 2 | 0

12. Primary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) up to 30 Days After the Second Vaccination
Description: A SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity.
Time Frame: From first vaccination (Day 1) up to 30 days post second vaccination (Day 91)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 101 | 97 | 100 | 101 | 101 | 100 | 103 | 100 | 101 | 101
Participants | 0 | 0 | 0 | 0 | 6 | 0 | 1 | 4 | 2 | 1 | 1 | 3 | 5 | 1

13. Primary Outcome: Number of Subjects With Any Potential Immune-mediated Diseases (pIMDs) up to 30 Days After the Second Vaccination (Part B Groups)
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: From first vaccination (Day 1) up to 30 days post second vaccination (Day 91)
Population: The analysis was performed on the Exposed Set that includes all subjects from Part B groups with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 101 | 97 | 100 | 101 | 101 | 100 | 103 | 100 | 101 | 101
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Subjects With Any SAEs, up the End of Follow-up Period (Month 14) - Part B Groups
Description: A SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 1 up to the end of follow-up period (Month 14)
Population: The analysis was performed on the Exposed Set that includes all subjects from Part B with at least one study vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 101 | 97 | 100 | 101 | 101 | 100 | 103 | 100 | 101 | 101
Participants | 13 | 3 | 5 | 8 | 6 | 11 | 9 | 5 | 9 | 9

15. Secondary Outcome: Number of Subjects Reporting pIMDs up to the End of Follow-up Period (Month 14) - Part B Groups
Description: as for outcome 13
Time Frame: From Day 1 up to the end of follow-up period (Month 14)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 101 | 97 | 100 | 101 | 101 | 100 | 103 | 100 | 101 | 101
Participants | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1

16. Secondary Outcome: Number of Subjects With at Least One RSV-confirmed Respiratory Tract Infection (RTI) Episode Post-vaccination Reported During RTI Surveillance - Part B Groups
Description: The number of subjects with at least one RTI case was provided by group. Reported categories are RSV+ (= RTI episode tested as RSV positive by quantitative reverse transcription polymerase chain reaction (qRT-PCR) on nasal/throat swab) and RSV- (= RTI episode tested as RSV negative by qRT-PCR on nasal/throat swab).
Time Frame: During the RSV season (from October 2019 to March 2020)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 101 | 97 | 100 | 101 | 101 | 100 | 103 | 100 | 101 | 101
Participants
  RSV+ | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
  RSV- | 19 | 12 | 20 | 14 | 17 | 22 | 20 | 16 | 13 | 11

17. Secondary Outcome: Humoral Immune Response With Respect to Components of the Investigational Vaccine in Terms of Neutralizing Antibody Titers Against RSV-serotype A
Description: Serological assays for the determination of functional antibodies against RSV-A were performed by neutralization assay. Anti RSV-A neutralizing antibody titers are given as geometric mean titers (GMTs) and expressed as Estimated Dose: serum dilution giving a 60% reduction of the signal compared to a control without serum (ED60).
Time Frame: At pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), on the day of second vaccination (Day 61) and 30 days post-Dose 2 (Day 91)
Population: The analysis was performed on the Per Protocol Set (PPS) that includes all subjects who receive the study treatment to which they are randomized and have post-vaccination data, minus subjects with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 11 | 11 | 12 | 12 | 101 | 96 | 99 | 100 | 101 | 100 | 102 | 100 | 101 | 100
Titers
  Day 1 | 1019 [634.6 to 1636.1] | 846.2 [481.7 to 1486.4] | 673.6 [325.3 to 1394.7] | 620.7 [365.1 to 1055.1] | 1015.5 [865 to 1192.2] | 1146.5 [931.6 to 1411] | 976.7 [837.7 to 1138.8] | 960.9 [801 to 1152.7] | 966.4 [822.9 to 1134.8] | 961.9 [809.5 to 1143] | 981.6 [832.7 to 1157.2] | 1023 [879.2 to 1190.2] | 1035.7 [864.5 to 1240.7] | 837.4 [701.3 to 999.9]
  Day 31: number analyzed (Participants) | 11 | 8 | 11 | 12 | 93 | 90 | 90 | 92 | 97 | 94 | 95 | 95 | 93 | 92
  Day 31 | 7658.4 [4329.7 to 13546.2] | 11741.8 [4883.6 to 28231.5] | 8136.9 [5066.1 to 13069.1] | 789.1 [518.6 to 1200.9] | 5422.6 [4395 to 6690.5] | 7371 [5922.5 to 9173.8] | 9403.1 [7471.2 to 11834.4] | 5258.5 [4351.8 to 6354.1] | 6509.4 [5306.8 to 7984.4] | 9350.9 [7606 to 11496.1] | 6026.1 [4960.9 to 7320.1] | 6899.5 [5767.8 to 8253.2] | 8527.7 [7107.9 to 10231] | 751.7 [625.2 to 903.9]
  Day 61: number analyzed (Participants) | 11 | 9 | 11 | 12 | 95 | 90 | 92 | 93 | 100 | 95 | 94 | 97 | 98 | 96
  Day 61 | 4659.8 [2090 to 10389.1] | 5895.8 [2791.9 to 12450.5] | 4761.5 [2687.7 to 8435.5] | 586.5 [333.1 to 1032.7] | 5657.9 [4736 to 6759.1] | 6490.8 [5190.3 to 8117.1] | 7907.4 [6253.9 to 9998.2] | 5019.4 [4281.5 to 5884.5] | 6201.9 [5106.3 to 7532.6] | 6681.7 [5498.4 to 8119.8] | 5048.9 [4184.4 to 6092] | 5902.1 [5023.4 to 6934.4] | 7201.4 [6000.4 to 8642.8] | 903.4 [750.8 to 1087.1]
  Day 91: number analyzed (Participants) | 11 | 8 | 11 | 12 | 88 | 84 | 87 | 84 | 91 | 87 | 85 | 93 | 92 | 93
  Day 91 | 6237.8 [3648.1 to 10665.9] | 5457.5 [2532.9 to 11758.7] | 3651 [1949.6 to 6837.2] | 787.9 [495.5 to 1252.6] | 3936.2 [3281.9 to 4720.9] | 5632.1 [4559.2 to 6957.5] | 5956.1 [4881.4 to 7267.4] | 3924.7 [3266 to 4716.2] | 4770 [3904.6 to 5827.4] | 5175.5 [4273.1 to 6268.5] | 4435.9 [3654.7 to 5384.1] | 4850.5 [4096.8 to 5742.8] | 5980.6 [4988 to 7170.7] | 772.4 [646.2 to 923.3]

18. Secondary Outcome: Humoral Immune Response With Respect to Components of the Investigational Vaccine in Terms of RSVPreF3-specific Immunoglobulin G (IgG) Antibody Concentrations
Description: The detection and the quantification of total IgG antibodies directed against RSVPreF3 in human serum samples were based on an indirect enzyme-linked immunosorbent assay (ELISA). Anti RSVPreF3 antibody concentration is given in geometric mean concentration (GMC) and is expressed in ELISA Laboratory Units per milliliter (ELU/mL).
Time Frame: as for outcome 17
Population: The analysis was performed on the PPS that includes all subjects who receive at least 1 dose of the study treatment to which they are randomized and have post-vaccination data, minus subjects with protocol deviations that lead to exclusion.
Measure: Geometric Mean (95% Confidence Interval); unit: ELU/mL
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 11 | 11 | 12 | 12 | 101 | 96 | 99 | 100 | 101 | 100 | 102 | 100 | 101 | 100
ELU/mL
  Day 1 | 8330.7 [5561.5 to 12478.9] | 7699.5 [5326 to 11130.8] | 7439.1 [5808.6 to 9527.2] | 6524.8 [4828.2 to 8817.6] | 7500.2 [6582.4 to 8545.9] | 7209.7 [6150.9 to 8450.7] | 7134.9 [6377.7 to 7982] | 6760.5 [5913.7 to 7728.5] | 7438 [6544.6 to 8453.4] | 6685.4 [5827 to 7670.4] | 7468.5 [6544 to 8523.5] | 7245.5 [6265.8 to 8378.3] | 6655.4 [5862.2 to 7555.9] | 6543.8 [5663 to 7561.6]
  Day 31: number analyzed (Participants) | 11 | 8 | 11 | 12 | 93 | 90 | 90 | 92 | 97 | 94 | 95 | 95 | 93 | 92
  Day 31 | 69843.3 [38345.8 to 127212.8] | 97848.5 [65057.1 to 147168] | 96645.4 [62880.7 to 148540.5] | 6601 [4888.4 to 8913.6] | 53994 [46566.7 to 62605.8] | 71618.4 [60729.6 to 84459.5] | 90933.2 [79096.2 to 104541.6] | 53598.9 [47062.7 to 61043] | 63823.4 [55601.6 to 73261] | 83462.5 [70906.1 to 98242.3] | 59026.1 [51236.4 to 68000] | 70524 [60825.4 to 81769.1] | 78831.2 [68382.5 to 90876.4] | 6593.4 [5672 to 7664.4]
  Day 61: number analyzed (Participants) | 11 | 9 | 11 | 12 | 95 | 90 | 93 | 93 | 100 | 95 | 94 | 97 | 98 | 96
  Day 61 | 50590.1 [27310.9 to 93711.7] | 58980.8 [38982.8 to 89237.7] | 56380.6 [38602.6 to 82346.1] | 6242.4 [4473 to 8711.7] | 47594.2 [41241.9 to 54924.8] | 56855.4 [47655.2 to 67831.7] | 70294.1 [61103.1 to 80867.5] | 41543.8 [36864.7 to 46816.8] | 51209.9 [44850.5 to 58470.9] | 62543.2 [52975.1 to 73839.3] | 45679.1 [39722.6 to 52528.7] | 54342.7 [47099 to 62700.5] | 61577.7 [53431.3 to 70966.1] | 6307.9 [5453.8 to 7295.9]
  Day 91: number analyzed (Participants) | 11 | 9 | 11 | 12 | 88 | 84 | 87 | 84 | 91 | 87 | 85 | 93 | 92 | 93
  Day 91 | 54900 [33635.4 to 89608.2] | 54884.7 [37768.6 to 79757.3] | 55444.4 [38128.6 to 80624] | 6246 [4375.8 to 8915.7] | 42523.7 [36905 to 48997.8] | 54711.2 [47013.5 to 63669.2] | 60955.2 [53029.7 to 70065.1] | 42504.6 [38044.3 to 47487.9] | 52846.4 [47105.8 to 59286.7] | 59624.5 [51680 to 68790.2] | 53779.9 [47588.5 to 60776.8] | 57314.9 [51038.1 to 64363.6] | 61433.7 [54066.2 to 69805] | 6748.7 [5804.1 to 7847.1]

19. Secondary Outcome: Descriptive Statistics of the Frequency of RSVPreF3 Specific Cluster of Differentiation 4+ (CD4+) T Cells Expressing at Least 2 Markers
Description: Among markers expressed were interleukin-2 (IL2), cluster of 40 ligand (CD40L), tumor necrosis factor alpha (TNF α) and interferon gamma (IFN γ), in vitro upon stimulation with RSVPreF3 peptide preparations. Reported statistics at each time point during which blood sample were collected for cell-mediated immunity, are geometric mean and inter-quartile range.
Time Frame: as for outcome 17
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: Cells per million CD4+ T Cells
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
Number analyzed (Participants) | 11 | 11 | 10 | 12 | 83 | 79 | 84 | 82 | 82 | 83 | 88 | 87 | 86 | 86
Cells per million CD4+ T Cells
  Day 1: number analyzed (Participants) | 11 | 11 | 10 | 11 | 82 | 77 | 84 | 82 | 82 | 83 | 80 | 87 | 86 | 84
  Day 1 | 400.0 [348 to 791] | 272.0 [163 to 570] | 317.5 [184 to 628] | 393.0 [333 to 680] | 208.5 [84 to 351] | 166.0 [75 to 291] | 225.5 [109 to 327] | 209.5 [127 to 338] | 188.0 [103 to 326] | 192.0 [67 to 381] | 187.5 [91 to 325.5] | 185.0 [82 to 294] | 206.0 [98 to 351] | 178.0 [100.5 to 293.5]
  Day 31: number analyzed (Participants) | 9 | 8 | 10 | 11 | 76 | 68 | 76 | 76 | 73 | 75 | 77 | 80 | 76 | 77
  Day 31 | 1649.0 [864 to 2604] | 2302.5 [1545 to 2725] | 1773.5 [1318 to 2124] | 303.0 [90 to 416] | 979.5 [639.5 to 1422.5] | 1089.5 [786 to 1812.5] | 1052.0 [674.5 to 1798] | 1594.0 [916 to 2360] | 1297.0 [881 to 2321] | 1466.0 [787 to 2116] | 1952.0 [1353 to 2953] | 1690.5 [1162.5 to 2691.5] | 1742.5 [1088 to 2360.5] | 176.0 [85 to 297]
  Day 61: number analyzed (Participants) | 10 | 8 | 9 | 11 | 83 | 79 | 82 | 77 | 81 | 79 | 88 | 86 | 84 | 86
  Day 61 | 1271.0 [519 to 1679] | 1515.0 [1129 to 2159] | 1066.0 [764 to 1502] | 263.0 [184 to 459] | 688.0 [430 to 1076] | 737.0 [437 to 1309] | 770.0 [479 to 1235] | 1086.0 [663 to 1621] | 1020.0 [603 to 1405] | 934.0 [598 to 1517] | 1228.5 [777.5 to 1832.5] | 1315.0 [887 to 1728] | 1078.0 [781 to 1631] | 183.0 [61 to 311]
  Day 91: number analyzed (Participants) | 10 | 8 | 9 | 12 | 79 | 79 | 82 | 74 | 80 | 78 | 78 | 83 | 80 | 84
  Day 91 | 1006.5 [872 to 1779] | 1221.0 [924 to 1518] | 1487.0 [1005 to 1664] | 374.5 [295 to 588] | 888.0 [650 to 1318] | 1034.0 [670 to 1598] | 1081.5 [769 to 1569] | 1732.0 [1163 to 2149] | 1603.5 [1087 to 2284] | 1496.0 [1179 to 2072] | 1966.0 [1339 to 2700] | 1558.0 [1263 to 2353] | 2096.5 [1441.5 to 2760.5] | 190.5 [100.5 to 308]

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected during the 7-day follow-up period after each vaccination. Unsolicited AEs were collected during the 30-day follow-up period after any vaccination. SAEs were collected during the whole study period, from Day 1 till Day 91 for Part A groups and till Month 14 for Part B groups.
Arm/Group | Low Dose_PLAIN_A Group | Medium Dose_PLAIN_A Group | High Dose_PLAIN_A Group | Placebo_A Group | Low Dose_PLAIN_B Group | Medium Dose_PLAIN_B Group | High Dose_PLAIN_B Group | Low Dose_AS01E_B Group | Medium Dose_AS01E_B Group | High Dose_AS01E_B Group | Low Dose_AS01B_B Group | Medium Dose_AS01B_B Group | High Dose_AS01B_B Group | Placebo_B Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/101 | 1/97 | 1/100 | 0/101 | 0/101 | 0/100 | 1/103 | 0/100 | 1/101 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 13/101 | 3/97 | 5/100 | 8/101 | 6/101 | 11/100 | 9/103 | 5/100 | 9/101 | 9/101
Other Adverse Events (participants affected / at risk) | 9/12 | 10/12 | 9/12 | 10/12 | 62/101 | 54/97 | 61/100 | 77/101 | 80/101 | 83/100 | 91/103 | 88/100 | 93/101 | 54/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose_PLAIN_A Group (N=12) | Medium Dose_PLAIN_A Group (N=12) | High Dose_PLAIN_A Group (N=12) | Placebo_A Group (N=12) | Low Dose_PLAIN_B Group (N=101) | Medium Dose_PLAIN_B Group (N=97) | High Dose_PLAIN_B Group (N=100) | Low Dose_AS01E_B Group (N=101) | Medium Dose_AS01E_B Group (N=101) | High Dose_AS01E_B Group (N=100) | Low Dose_AS01B_B Group (N=103) | Medium Dose_AS01B_B Group (N=100) | High Dose_AS01B_B Group (N=101) | Placebo_B Group (N=101)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal cord infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hormone receptor positive breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung carcinoma cell type unspecified stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sarcoma uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose_PLAIN_A Group (N=12) | Medium Dose_PLAIN_A Group (N=12) | High Dose_PLAIN_A Group (N=12) | Placebo_A Group (N=12) | Low Dose_PLAIN_B Group (N=101) | Medium Dose_PLAIN_B Group (N=97) | High Dose_PLAIN_B Group (N=100) | Low Dose_AS01E_B Group (N=101) | Medium Dose_AS01E_B Group (N=101) | High Dose_AS01E_B Group (N=100) | Low Dose_AS01B_B Group (N=103) | Medium Dose_AS01B_B Group (N=100) | High Dose_AS01B_B Group (N=101) | Placebo_B Group (N=101)
Injection site pain (General disorders) | 6 (6) | 9 (14) | 8 (14) | 1 (1) | 23 (27) | 19 (23) | 31 (37) | 60 (89) | 63 (105) | 65 (103) | 81 (136) | 78 (120) | 82 (137) | 8 (8)
Fatigue (General disorders) | 5 (7) | 5 (7) | 4 (5) | 7 (11) | 29 (39) | 20 (22) | 29 (37) | 41 (51) | 39 (51) | 36 (46) | 45 (66) | 47 (64) | 53 (83) | 24 (32)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 11 (15) | 7 (8) | 6 (7) | 21 (26) | 19 (20) | 19 (25) | 3 (3)
Injection site swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 8 (10) | 9 (10) | 11 (12) | 17 (20) | 9 (14) | 14 (19) | 0 (0)
Hangover (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 4 (4) | 2 (2) | 6 (7) | 8 (9) | 6 (6) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 2 (2)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site movement impairment (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site paraesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 9 (10) | 8 (10) | 4 (4) | 14 (17) | 19 (23) | 18 (19) | 28 (37) | 19 (23) | 24 (31) | 11 (14)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 6 (7) | 5 (6) | 14 (17) | 12 (17) | 15 (17) | 28 (39) | 22 (24) | 32 (36) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 4 (4) | 3 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (2) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (4) | 5 (6) | 5 (6) | 5 (7) | 16 (19) | 14 (18) | 17 (21) | 28 (36) | 25 (32) | 24 (29) | 45 (61) | 38 (54) | 38 (48) | 13 (17)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (3) | 3 (3) | 11 (13) | 9 (10) | 14 (17) | 13 (15) | 11 (13) | 15 (16) | 18 (24) | 12 (15) | 19 (22) | 13 (16)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palatal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic cyst (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 7 (8) | 9 (9) | 14 (16) | 24 (33) | 20 (29) | 24 (30) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 3 (3) | 4 (4) | 3 (3) | 4 (5) | 3 (3) | 4 (5) | 2 (2) | 6 (6) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sialoadenitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulpitis dental (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 3 (3) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal discharge discolouration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart rate irregular (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoferritinaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reaction to preservatives (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermoid cyst (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/90/NCT03814590/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/90/NCT03814590/SAP_001.pdf